CLINICAL TRIAL: NCT01908829
Title: A Randomized, Double-Blind, Multi-Centre Study to Evaluate the Efficacy and Safety of Adding Mirabegron to Solifenacin in Incontinent OAB Subjects Who Have Received Solifenacin for 4 Weeks and Warrant Additional Relief for Their OAB Symptoms
Brief Title: A Trial Comparing Combination Treatment (Solifenacin Plus Mirabegron) With One Treatment Alone (Solifenacin)
Acronym: BESIDE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Europe Ltd. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 905-EC-012; 2012-005401-41 (EudraCT Number)
Record Dates: First submitted 2013-07-24; First posted 2013-07-26 (Estimated); Results first posted 2017-10-09 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Urinary Bladder Diseases; Urinary Bladder Overactive; Urologic Diseases
Keywords: Vesitrim; Betanis; Urgency; Frequency; Mirabegron; YM178; Betmiga; Vesicare; Micturition; YM905; Solifenacin; Urinary incontinence; Overactive Bladder (OAB); Myrbetriq; Vesikur; Urgency incontinence
MeSH Terms: conditions — Urinary Bladder Diseases; Urinary Bladder, Overactive; Urologic Diseases; Urinary Incontinence | interventions — mirabegron; Solifenacin Succinate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Combination (solifenacin + mirabegron) (Experimental): Participants received solifenacin 5 mg, mirabegron 25 mg and solifenacin 10 mg matching placebo once daily for the first 4 weeks of double-blind period. For the last 8 weeks of the double-blind treatment period, the 25 mg mirabegron tablet was replaced by a 50 mg mirabegron tablet. Placebo was given for the 2 week single-blind safety follow-up period.
  Interventions: Drug: mirabegron 25 mg; Drug: mirabegron 50 mg; Drug: solifenacin 5 mg; Drug: solifenacin 10 mg matching placebo
- Solifenacin 5 mg (Active Comparator): Participants received solifenacin 5 mg, mirabegron 25 mg matching placebo and solifenacin 10 mg matching placebo once daily. For the last 8 weeks of the double-blind treatment period, the 25 mg mirabegron matching placebo tablet was replaced by a 50 mg mirabegron matching placebo tablet (to maintain the blind). Placebo was given for the 2 week single-blind safety follow-up period
  Interventions: Drug: solifenacin 5 mg; Drug: mirabegron 25 mg matching placebo; Drug: mirabegron 50 mg matching placebo; Drug: solifenacin 10 mg matching placebo
- Solifenacin 10 mg (Active Comparator): Participants received solifenacin 5 mg matching placebo, mirabegron 25 mg matching placebo and solifenacin 10 mg once daily. For the last 8 weeks of the double-blind treatment period, the 25 mg mirabegron matching placebo tablet was replaced by a 50 mg mirabegron matching placebo tablet (to maintain the blind). Placebo was given for the 2 week single-blind safety follow-up period.
  Interventions: Drug: solifenacin 10 mg; Drug: mirabegron 25 mg matching placebo; Drug: mirabegron 50 mg matching placebo; Drug: solifenacin 5 mg matching placebo

INTERVENTIONS:
Drug: mirabegron 25 mg — Mirabegron was supplied as the marketed formulation in the 25 mg OCAS (Oral Controlled Absorption System) modified release tablets. Medication was taken orally with a glass of water, with or without food.
  Other Names: Betmiga; Myrbetriq; YM178; Betanis
  Arms: Combination (solifenacin + mirabegron)
Drug: mirabegron 50 mg — Mirabegron was supplied as the marketed formulation in the 50 mg OCAS (Oral Controlled Absorption System) modified release tablets. Medication was taken orally with a glass of water, with or without food.
  Other Names: YM905; Vesitrim; Vesikur; Vesicare
  Arms: Combination (solifenacin + mirabegron)
Drug: solifenacin 5 mg — Solifenacin was provided as the marketed formulation in the 5 mg strength. Medication was taken orally with a glass of water, with or without food.
  Other Names: Vesicare; Vesitrim; YM905; Vesikur
  Arms: Combination (solifenacin + mirabegron); Solifenacin 5 mg
Drug: solifenacin 10 mg — Solifenacin was provided as the marketed formulation in the 10 mg strength. Medication was taken orally with a glass of water, with or without food.
  Other Names: Vesicare; Vesitrim; YM905; Vesikur
  Arms: Solifenacin 10 mg
Drug: mirabegron 25 mg matching placebo — Matching placebo of mirabegron OCAS 25 mg tablets was supplied. Medication was taken orally with a glass of water, with or without food.
  Arms: Solifenacin 10 mg; Solifenacin 5 mg
Drug: mirabegron 50 mg matching placebo — Matching placebo of mirabegron OCAS 50 mg tablets was supplied. Medication was taken orally with a glass of water, with or without food.
  Arms: Solifenacin 10 mg; Solifenacin 5 mg
Drug: solifenacin 5 mg matching placebo — Matching placebo of solifenacin succinate 5 mg tablets was supplied. Medication was taken orally with a glass of water, with or without food.
  Arms: Solifenacin 10 mg
Drug: solifenacin 10 mg matching placebo — Matching placebo of solifenacin succinate 10 mg tablets was supplied. Medication was taken orally with a glass of water, with or without food.
  Arms: Combination (solifenacin + mirabegron); Solifenacin 5 mg

SUMMARY:
The purpose of this study was to see if adding a new type of medication recently approved to treat overactive bladder (mirabegron) to an antimuscarinic treatment (solifenacin) would be more effective in controlling incontinence than when using the antimuscarinic treatment alone.

ELIGIBILITY:
Inclusion Criteria:

* Main Inclusion at Screening:

  1. Subject has symptoms of OAB (urinary frequency and urgency with urgency incontinence) for >= 3 months prior to the screening visit
  2. Subject is willing and able to complete the micturition diary and questionnaires correctly, including collection and measurement of urine output for 3 days prior to each visit;
  3. Subject has symptoms of "wet" OAB (urinary frequency and urgency with incontinence or mixed incontinence with predominant urgency incontinence), and reports an average of at least 2 incontinence episodes per day.
* Main Inclusion at Run-in (Visit 2):

  1. Subject experiences on average at least 1 episode of urgency (grade 3 or 4) with or without incontinence per 24-hour period during the 3-day micturition diary period.
  2. Subject experiences on average at least 2 incontinence episodes per 24-hour period during the 3-day micturition diary period.
  3. Subject experiences on average at least 8 micturitions (excluding incontinence episodes) per 24-hour period during the 3-day micturition diary period.
* Main Inclusion at Randomization (Visit 3):

  1. Subject experiences at least 1 incontinence episode during the 3-day micturition diary period and wishes to increase their treatment for OAB symptoms.

Exclusion Criteria:

* Main Exclusion at Screening:

  1. Subject in the opinion of the investigator has clinically significant Bladder Outlet Obstruction (BOO).
  2. Subject has significant Post-void residual (PVR) volume (PVR > 150 ml).
  3. Subject has significant stress incontinence or mixed stress/urgency incontinence where stress is the predominant factor as determined by the investigator
  4. Subject has an indwelling catheter or practices intermittent self catheterization.
  5. Subject has evidence of a UTI.
  6. Subject has chronic inflammation such as interstitial cystitis, bladder stones, previous pelvic radiation therapy, or previous or current malignant disease of the pelvic organs
  7. Subject has moderate to severe hepatic impairment
  8. Subject has severe renal impairment or End Stage Renal disease
  9. Subject has a clinically significant abnormal Electrocardiogram (ECG)
  10. Subject has a concurrent malignancy or history of cancer (except noninvasive skin cancer) within the last 5 years prior to screening.
  11. Subject has a QTcF interval > 450 ms for males or > 470 ms for females or is at risk of QT prolongation (e.g., family history of long QT syndrome, hypokalaemia).
  12. Subject has received intravesical treatment in the past 12 months with e.g., botulinum toxin, resiniferatoxin, capsaicin.
  13. Subject has severe uncontrolled hypertension, which is defined as a sitting average systolic blood pressure ≥ 180 mmHg and/or average diastolic blood pressure ≥ 110 mmHg.
* Main Exclusion at Randomization (visit 3):

  1. Subject has achieved 100% continence from Visit 2 to Visit 3 (no incontinence episodes are recorded in the 3 day diary administered for 3 days prior to Visit 3).
  2. Subject does not desire an increase in study medication.
  3. Subject has an average total daily urine volume > 3000ml as recorded in the micturition diary.
  4. Subject has severe uncontrolled hypertension, which is defined as a sitting average systolic blood pressure ≥ 180 mmHg and/or average diastolic blood pressure ≥ 110 mmHg.
  5. Subject has a clinically significant abnormal ECG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2174 (Actual)
Dates: Start 2013-07-10 (Actual); Primary Completion 2014-11-24 (Actual); Study Completion 2014-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Manager, Study Director — Astellas Pharma Europe Ltd.
Locations (219):
- United States (36):
  - Genova Clinical Research, Tucson, Arizona
  - Associated Pharmaceutical Research Center, Inc., Buena Park, California
  - The American Institute of Research, Los Angeles, California
  - Bayview Research Group, Valley Village, California
  - Meridien Research, Brooksville, Florida
  - Innovative Research of West FL, Clearwater, Florida
  - Best Quality Research Inc., Hialeah, Florida
  - Palmetto Professional Research, Hialeah, Florida
  - Urology Center of Central Florida, Kissimmee, Florida
  - Meridien Research, Tampa, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Private Practice, West Palm Beach, Florida
  - Meridian Clinical Research, LLC, Savannah, Georgia
  - Herman Clinical Research, Suwanee, Georgia
  - North Idaho Urology, Coeur d'Alene, Idaho
  - First Urology, PSC, Jeffersonville, Indiana
  - Deaconess Gateway Health Center, Newburgh, Indiana
  - MedStar Health Research Institute, Hyattsville, Maryland
  - Bay State Clinical Trials, Inc., Watertown, Massachusetts
  - Beyer Research, Kalamazoo, Michigan
  - Quality Clinical Research, Omaha, Nebraska
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - Brooklyn Urology Research Group, Brooklyn, New York
  - Advanced Urology Centers of New York, Garden City, New York
  - Premier Medical Group of the Hudson Valley PC, Kingston, New York
  - Premier Medical Group of the Hudson Valley PC, Poughkeepsie, New York
  - PMG Research of Raleigh, dba PMG Research of Cary, Cary, North Carolina
  - Alliance Urology Specialists, Greensboro, North Carolina
  - Wake Research Associates LLC, Raleigh, North Carolina
  - PMG Research of Winston-Salem, LLC, Winston-Salem, North Carolina
  - The Urology Group, Cincinnati, Ohio
  - Providence Health Partners, Dayton, Ohio
  - The Clinical Trial Center, Jenkintown, Pennsylvania
  - Health Concepts, Rapid City, South Dakota
  - Jean Brown Research, Salt Lake City, Utah
  - Alexandria Clinical Research, Alexandria, Virginia
- Armenia (3):
  - Site: 37402, Yerevan
  - Site: 37403, Yerevan
  - Site: 37405, Yerevan
- Australia (3):
  - Site: 61006, Adelaide
  - Site: 61001, Kogarah, Sydney
  - Site: 61016, Victoria
- Austria (11):
  - Site: 43008, Graz
  - Site: 43001, Innsbruck
  - Site: 43006, Innsbruck
  - Site: 43007, Linz
  - Site: 43002, Vienna
  - Site: 43004, Vienna
  - Site: 43005, Vienna
  - Site: 43010, Vienna
  - Site: 43011, Vienna
  - Site: 43012, Vienna
  - Site: 43003, Wels
- Belgium (8):
  - Site: 32007, Anderlecht
  - Site: 32013, Deurne
  - Site: 32009, Edegem
  - Site: 32003, Ghent
  - Site: 32005, Ghent
  - Site: 32015, Kortrijk
  - Site: 32008, Liège
  - Site: 32014, Roeselare
- Canada (12):
  - Site: 15001, Barrie
  - Site: 15009, Bathurst
  - Site: 15006, Brampton
  - Site: 15015, Granby
  - Site: 15014, Kelowna
  - Site: 15007, Kitchener
  - Site: 15019, Sherbrooke
  - Site: 15012, Toronto
  - Site: 15013, Toronto
  - Site: 15016, Victoria
  - Site: 15047, Victoria
  - Site: 15018, Victoriaville
- Czechia (10):
  - Site: 42015, Brno
  - Site: 42020, Mělník
  - Site: 42018, Náchod
  - Site: 42004, Pilsen
  - Site: 42021, Pilsen
  - Site: 42007, Prague
  - Site: 42008, Prague
  - Site: 42016, Prague
  - Site: 42017, Prague
  - Site: 42022, Prague
- Denmark (4):
  - Site: 45008, Aarhus N
  - Site: 45003, Frederiksberg
  - Site: 45009, Herlev
  - Site: 45011, Odense C
- Finland (2):
  - Site: 35804, Helsinki (hus)
  - Site: 35805, Tampere
- France (2):
  - Site: 33018, Bordeaux
  - Site: 33017, Marseille
- Site: 99502, Tbilisi, Georgia
- Germany (11):
  - Site: 49008, Bad Ems
  - Site: 49022, Berlin
  - Site: 49003, Eisleben Lutherstadt
  - Site: 49021, Hagenow
  - Site: 49011, Halle
  - Site: 49004, Hamburg
  - Site: 49018, Henningsdorf
  - Site: 49009, Hettstedt
  - Site: 49017, Koblenz
  - Site: 49020, Reutlingen
  - Site: 49014, Sangerhausen
- Greece (3):
  - Site: 30001, Athens
  - Site: 30005, Heraklion, Crete
  - Site: 30002, Pátrai
- Hungary (5):
  - Site: 36003, Csongrád
  - Site: 36011, Hajdúszoboszló
  - Site: 36002, Nyíregyháza
  - Site: 36008, Salgótarján
  - Site: 36009, Szekszárd
- Ireland (8):
  - Site: 35303, Cork
  - Site: 35301, Dublin
  - Site: 35309, Dublin
  - Site: 35310, Dublin
  - Site: 35306, Limerick
  - Site: 35313, Mullingar
  - Site: 35304, Tralee
  - Site: 35305, Waterford
- Israel (6):
  - Site: 97201, Haifa
  - Site: 97202, Jerusalem
  - Site: 97207, Kfar Saba
  - Site: 97203, Petah Tikva
  - Site: 97205, Petah Tikva
  - Site: 97206, Tel Litwinsky
- Italy (6):
  - Site: 39007, Avellino
  - Site: 39002, Cantanzaro
  - Site: 39010, Florence
  - Site: 39006, Perugia
  - Site: 39013, Treviglio (BG)
  - Site: 39009, Varese
- Site: 96101, Beirut, Lebanon
- Site: 31008, Amsterdam, Netherlands
- Norway (3):
  - Site: 47005, Bekkestua
  - Site: 47003, Trondheim
  - Site: 47002, Tønsberg
- Poland (6):
  - Site: 48002, Kolbuszowa Dolna
  - Site: 48006, Krakow
  - Site: 48010, Lublin
  - Site: 48005, Piaseczno
  - Site: 48001, Warsaw
  - Site: 48008, Warsaw
- Portugal (6):
  - Site: 35104, Lisbon
  - Site: 35105, Lisbon
  - Site: 35102, Matosinhos Municipality
  - Site: 35103, Porto
  - Site: 35101, Setúbal
  - Site: 35106, Tomar
- Romania (7):
  - Site: 40016, Bucharest
  - Site: 40018, Bucharest
  - Site: 40012, Craiova
  - Site: 40019, Craiova
  - Site: 40003, Judetul Ilfov
  - Site: 40017, Oradea
  - Site: 40020, Timișoara
- Russia (14):
  - Site: 70003, Moscow
  - Site: 70004, Moscow
  - Site: 70005, Moscow
  - Site: 70008, Moscow
  - Site: 70010, Moscow
  - Site: 70011, Moscow
  - Site: 70012, Moscow
  - Site: 70024, Moscow
  - Site: 70013, Rostove-on-Don
  - Site: 70002, Saint Petersburg
  - Site: 70006, Saint Petersburg
  - Site: 70007, Saint Petersburg
  - Site: 70009, Saint Petersburg
  - Site: 70025, Saratov
- Slovakia (7):
  - Site: 42110, Bratislava
  - Site: 42114, Košice
  - Site: 42113, Michalovce
  - Site: 42111, Nové Zámky
  - Site: 42112, Piešťany
  - Site: 42108, Poprad
  - Site: 42109, Žilina
- Slovenia (4):
  - Site: 38601, Ljubljana
  - Site: 38606, Maribor
  - Site: 38607, Maribor
  - Site: 38610, Ptuj
- Spain (12):
  - Site: 34012, Barcelona
  - Site: 34016, Bilbao
  - Site: 34013, Donostia / San Sebastian
  - Site: 34001, Getafe (Madrid)
  - Site: 34004, Madrid
  - Site: 34015, Madrid
  - Site: 34023, Mendaro
  - Site: 34021, Miranda de Ebro
  - Site: 34018, San Sebastián de los Reyes
  - Site: 34007, Seville
  - Site: 34020, Seville
  - Site: 34014, Vigo
- Sweden (6):
  - Site: 46004, Halmstad
  - Site: 46013, Lund
  - Site: 46014, Norrtälje
  - Site: 46001, Stockholm
  - Site: 46012, Stockholm
  - Site: 46015, Umeå
- Switzerland (2):
  - Site: 41008, Baden
  - Site: 41001, Frauenfeld
- Turkey (Türkiye) (7):
  - Site: 90005, Ankara
  - Site: 90008, Ankara
  - Site: 90002, Izmir
  - Site: 90003, Izmir
  - Site: 90007, Kocaeli
  - Site: 90004, Manisa
  - Site: 90006, Sivas
- United Kingdom (12):
  - Site: 44007, Bristol
  - Site: 44012, Cambridge
  - Site: 44015, Cheltenham
  - Site: 44019, Coventry
  - Site: 44009, Garston
  - Site: 44016, Kings Lynn
  - Site: 44017, London
  - Site: 44018, Northampton
  - Site: 44010, Nottingham
  - Site: 44008, Plymouth
  - Site: 44013, Taunton
  - Site: 44011, West Yorkshire

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Gibson W, MacDiarmid S, Huang M, Siddiqui E, Stolzel M, Choudhury N, Drake MJ. Treating Overactive Bladder in Older Patients with a Combination of Mirabegron and Solifenacin: A Prespecified Analysis from the BESIDE Study. Eur Urol Focus. 2017 Dec;3(6):629-638. doi: 10.1016/j.euf.2017.08.008. Epub 2017 Sep 12. PMID 28916436
- [Derived] Drake MJ, Chapple C, Esen AA, Athanasiou S, Cambronero J, Mitcheson D, Herschorn S, Saleem T, Huang M, Siddiqui E, Stolzel M, Herholdt C, MacDiarmid S; BESIDE study investigators. Efficacy and Safety of Mirabegron Add-on Therapy to Solifenacin in Incontinent Overactive Bladder Patients with an Inadequate Response to Initial 4-Week Solifenacin Monotherapy: A Randomised Double-blind Multicentre Phase 3B Study (BESIDE). Eur Urol. 2016 Jul;70(1):136-145. doi: 10.1016/j.eururo.2016.02.030. Epub 2016 Mar 8. PMID 26965560
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=247

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study was conducted at 281 centers globally. Randomization was stratified by sex, age group (< 65, ≥ 65 years), 4-week incontinence episode reduction group (< 50%, ≥ 50%) and geographic region.
Pre-assignment Details: Participants who met the screening inclusion/exclusion criteria went through a two week wash-out period and maintained a micturition diary during that the wash-out period. A total of 3815 participants were screened of which 2401 participants received solifenacin 5 mg run-in medication. A total of 2174 participants were randomized.
Period: Overall Study
Arm/Group | Combination (Solifenacin + Mirabegron) | Solifenacin 5 mg | Solifenacin 10 mg
Started | 727 | 728 | 719
Treated With Double-blind Drug | 725 | 728 | 719
Completed | 678 | 679 | 680
Not Completed | 49 | 49 | 39
Not completed — Adverse Event | 13 | 11 | 13
Not completed — Lost to Follow-up | 4 | 2 | 1
Not completed — Randomized no double-blind drug received | 1 | 0 | 1
Not completed — Discontinued (no EoT page) | 2 | 0 | 0
Not completed — Miscellaneous | 0 | 2 | 0
Not completed — Protocol Violation | 2 | 2 | 0
Not completed — Lack of Efficacy | 1 | 3 | 2
Not completed — Withdrawal by Subject | 26 | 29 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Combination (Solifenacin + Mirabegron) | Solifenacin 5 mg | Solifenacin 10 mg | Total
Number analyzed (Participants) | 727 | 728 | 719 | 2174
Age, Continuous [Mean (Standard Deviation); unit: Year] | 58.2 (13.1) | 56.9 (13.5) | 57.4 (13.2) | 57.5 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 604 | 604 | 600 | 1808
  Male | 123 | 124 | 119 | 366

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to End of Treatment (EoT) in Mean Number of Incontinence Episodes Per 24 Hours
Description: The mean number of incontinence episodes (complaint of any involuntary leakage of urine) per day was derived from number of incontinence episodes recorded on valid diary days during the 3-day micturition diary period divided by the number of valid diary days during the 3-day micturition diary period. The analysis population consisted of the Full Analysis Set (FAS) which comprised of all the Randomized Analysis Set's (RAS) participants who met the following criteria: took at least 1 dose of double-blind study drug after randomization, reported at least 1 micturition in the baseline diary & at least 1 micturition postbaseline & reported at least 1 incontinence episode in the baseline diary. For participants who withdrew before EoT (week 12) and have no measurement available for that diary period, the Last Observation Carried Forward (LOCF) value during the double-blind study period was used as EoT value to derive the primary variable.
Time Frame: Baseline and end of treatment (up to 12 weeks)
Population: The analysis population consisted of the FAS. LOCF was used for EoT.
Measure: Least Squares Mean (Standard Error); unit: incontinence episodes
Arm/Group | Combination (Solifenacin + Mirabegron) | Solifenacin 5 mg | Solifenacin 10 mg
Number analyzed (Participants) | 706 | 704 | 697
incontinence episodes | -1.8 (0.08) | -1.53 (0.08) | -1.67 (0.08)
Statistical Analysis 1: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; Differences of adjusted means were calculated by subtracting adjusted mean of solifenacin monotherapy groups from adjusted mean of combination group based on ANCOVA model. Means (LS means) and 95% Confidence Intervals (CIs) are from an ANCOVA model with sex, age group (< 65, ≥ 65 years), geographic region, and 4-week incontinence episode reduction group as fixed factors and mean number of incontinence episodes per 24 hours at baseline as a covariate; Test type: Superiority; p = 0.001, stratified rank ANCOVA — P values for pairwise comparisons were from the stratified rank ANCOVA model. P < 0.05 indicated superiority in favor of treatment group with the largest improvement; Least Squares (LS) Means = -0.26, 95% CI 2-sided [-0.47 to -0.05], Standard Error of Mean 0.11

2. Secondary Outcome: Change From Baseline to Weeks 4, 8 & 12 in Mean Number of Incontinence Episodes Per 24 Hours
Description: The mean number of incontinence episodes (complaint of any involuntary leakage of urine) per day was derived from number of incontinence episodes recorded on valid diary days during the 3-day micturition diary period divided by the number of valid diary days during the 3-day micturition diary period.
Time Frame: Baseline and weeks 4, 8 & 12
Population: The analysis population consisted of the FAS with data available at each time point.
Measure: Least Squares Mean (Standard Error); unit: incontinence episodes
Arm/Group | Combination (Solifenacin + Mirabegron) | Solifenacin 5 mg | Solifenacin 10 mg
Number analyzed (Participants) | 707 | 705 | 698
incontinence episodes
  Week 4: number analyzed (Participants) | 690 | 690 | 679
  Week 4 | -1.24 (0.07) | -0.91 (0.07) | -1.12 (0.07)
  Week 8: number analyzed (Participants) | 661 | 674 | 673
  Week 8 | -1.68 (0.07) | -1.29 (0.07) | -1.49 (0.07)
  Week 12: number analyzed (Participants) | 653 | 645 | 664
  Week 12 | -1.81 (0.08) | -1.57 (0.08) | -1.67 (0.08)
Statistical Analysis 1: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; Week 4 differences of adjusted means were calculated by subtracting adjusted mean of solifenacin monotherapy groups from adjusted mean of combination group based on ANCOVA model. Means (LS means) and 95% CIs are from an ANCOVA model with sex, age group (< 65, ≥ 65 years), geographic region, and 4-week incontinence episode reduction group as fixed factors and mean number of incontinence episodes per 24 hours at baseline as a covariate; Test type: Superiority; p < 0.001, stratified rank ANCOVA — P values for pairwise comparisons are from the stratified rank ANCOVA model. P < 0.05 indicates superiority in favor of treatment group with the largest improvement; LS Means = -0.33, 95% CI 2-sided [-0.52 to -0.14], Standard Error of Mean 0.10
Statistical Analysis 2: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; Week 8 differences of adjusted means were calculated by subtracting adjusted mean of solifenacin monotherapy groups from adjusted mean of combination group based on ANCOVA model. Means (LS means) and 95% CIs are from an ANCOVA model with sex, age group (< 65, ≥ 65 years), geographic region, and 4-week incontinence episode reduction group as fixed factors and mean number of incontinence episodes per 24 hours at baseline as a covariate; Test type: Superiority; p < 0.001, stratified rank ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Means = -0.39, 95% CI 2-sided [-0.60 to -0.18], Standard Error of Mean 0.10
Statistical Analysis 3: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; Week 12 differences of adjusted means were calculated by subtracting adjusted mean of solifenacin monotherapy groups from adjusted mean of combination group based on ANCOVA model. Means (LS means) and 95% CIs are from an ANCOVA model with sex, age group (< 65, ≥ 65 years), geographic region, and 4-week incontinence episode reduction group as fixed factors and mean number of incontinence episodes per 24 hours at baseline as a covariate; Test type: Superiority; p = 0.001, stratified rank ANCOVA — P-values for pairwise comparisons are from the stratified rank ANCOVA model. p<0.05 indicates superiority in favor of treatment group with the largest improvement; LS Means = -0.25, 95% CI 2-sided [-0.46 to -0.03], Standard Error of Mean 0.11

3. Secondary Outcome: Change From Baseline in Mean Number of Micturitions Per 24 Hours
Description: The average number of micturitions (voluntary urinations (excluding incontinence only episodes)) per 24 hours was derived from number of micturitions recorded on valid diary days during the 3-day micturition diary period divided by the number of valid diary days during the 3-day micturition diary period (excluding incontinence only episodes).
Time Frame: Baseline and weeks 4, 8 & 12
Population: LOCF was used for EoT. The analysis population consisted of the FAS with data available at each time point.
Measure: Least Squares Mean (Standard Error); unit: micturitions
Arm/Group | Combination (Solifenacin + Mirabegron) | Solifenacin 5 mg | Solifenacin 10 mg
Number analyzed (Participants) | 707 | 705 | 698
micturitions
  Week 4: number analyzed (Participants) | 690 | 690 | 679
  Week 4 | -0.95 (0.07) | -0.69 (0.07) | -0.79 (0.07)
  Week 8: number analyzed (Participants) | 661 | 674 | 673
  Week 8 | -1.36 (0.08) | -0.94 (0.08) | -1.00 (0.08)
  Week 12: number analyzed (Participants) | 653 | 645 | 664
  Week 12 | -1.63 (0.08) | -1.16 (0.09) | -1.11 (0.08)
  EoT: number analyzed (Participants) | 706 | 704 | 697
  EoT | -1.59 (0.08) | -1.14 (0.08) | -1.12 (0.08)
Statistical Analysis 1: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; Week 4 adjusted change from baseline values as well as 95% CIs and p-value were generated from an ANCOVA model with treatment group, sex, age group (<65, >=65 years), 4-week incontinence reduction group and geographic region as fixed factors and baseline value as a covariate. Differences of adjusted means were calculated by subtracting adjusted mean of solifenacin monotherapy groups from adjusted mean of combination group; Test type: Superiority; p = 0.010, ANCOVA — P-values for pairwise comparisons are from the ANCOVA model described above. p<0.05 indicates superiority in favor of treatment group with the largest improvement; LS Means = -0.26, 95% CI 2-sided [-0.47 to -0.06], Standard Error of Mean 0.10
Statistical Analysis 2: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; Week 8 adjusted change from baseline values as well as 95% CIs and p-value were generated from an ANCOVA model with treatment group, sex, age group (<65, >=65 years), 4-week incontinence reduction group and geographic region as fixed factors and baseline value as a covariate. Differences of adjusted means were calculated by subtracting adjusted mean of solifenacin monotherapy groups from adjusted mean of combination group; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS Means = -0.42, 95% CI 2-sided [-0.65 to -0.19], Standard Error of Mean 0.12
Statistical Analysis 3: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; Week 12 adjusted change from baseline values as well as 95% CIs and p-value were generated from an ANCOVA model with treatment group, sex, age group (<65, >=65 years), 4-week incontinence reduction group and geographic region as fixed factors and baseline value as a covariate. Differences of adjusted means were calculated by subtracting adjusted mean of solifenacin monotherapy groups from adjusted mean of combination group; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS Means = -0.47, 95% CI 2-sided [-0.70 to -0.23], Standard Error of Mean 0.12
Statistical Analysis 4: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; EoT adjusted change from baseline values as well as 95% CIs and p-value were generated from an ANCOVA model with treatment group, sex, age group (<65, >=65 years), 4-week incontinence reduction group and geographic region as fixed factors and baseline value as a covariate. Differences of adjusted means were calculated by subtracting adjusted mean of solifenacin monotherapy groups from adjusted mean of combination group; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS Means = -0.45, 95% CI 2-sided [-0.67 to -0.22], Standard Error of Mean 0.12

4. Secondary Outcome: Number of Incontinence Episodes Reported During the 3-Day Diary
Description: The number of incontinence episodes (complaint of any involuntary leakage of urine) per day was derived from total number of incontinence episodes on valid diary days recorded during the 3-day micturition diary period.
Time Frame: Weeks 4, 8 and 12
Population: LOCF was used for EoT. The analysis population consisted of the FAS with data available at each time point.
Measure: Mean (Standard Error); unit: incontinence episodes
Arm/Group | Combination (Solifenacin + Mirabegron) | Solifenacin 5 mg | Solifenacin 10 mg
Number analyzed (Participants) | 707 | 705 | 698
incontinence episodes
  Week 4: number analyzed (Participants) | 690 | 690 | 679
  Week 4 | 5.81 (0.30) | 6.68 (0.31) | 6.41 (0.33)
  Week 8: number analyzed (Participants) | 661 | 674 | 673
  Week 8 | 4.55 (0.30) | 5.43 (0.30) | 5.28 (0.32)
  Week 12: number analyzed (Participants) | 653 | 645 | 664
  Week 12 | 4.03 (0.29) | 4.56 (0.28) | 4.62 (0.31)
  EoT: number analyzed (Participants) | 706 | 704 | 697
  EoT | 4.25 (0.29) | 4.87 (0.28) | 4.72 (0.31)
Statistical Analysis 1: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; Week 4 rate ratio, 95% CIs, & p-value for number of incontinence episodes (IEs) during Week 4 3-day diary between combination & solifenacin treatment was calculated from Mixed Effects Poisson (negative binomial) regression model including treatment group, sex, age group (<65, >=65 years), geographic region & 4-week IE reduction group as factors, log of (number of IEs/valid diary days) at baseline as covariate & log of number of valid diary days as the offset variable; Test type: Superiority; p = 0.005, Mixed Effects Poisson — p<0.05 indicates superiority in favor of treatment group with lowest rate of incontinence episodes; Rate Ratio = 0.87, 95% CI 2-sided [0.79 to 0.96], Standard Error of Mean 0.05
Statistical Analysis 2: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; Week 8 rate ratio, 95% CIs, & p-value for number of incontinence episodes (IEs) during Week 8 3-day diary between combination & solifenacin treatment was calculated from Mixed Effects Poisson (negative binomial) regression model including treatment group, sex, age group (<65, >=65 years), geographic region & 4-week IE reduction group as factors, log of (number of IEs/valid diary days) at baseline as covariate & log of number of valid diary days as the offset variable; Test type: Superiority; p < 0.001, Mixed Effects Poisson — p<0.05 indicates superiority in favor of treatment group with lowest rate of incontinence episodes; Rate Ratio = 0.75, 95% CI 2-sided [0.66 to 0.86], Standard Error of Mean 0.07
Statistical Analysis 3: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; Week 12 rate ratio, 95% CIs, & p-value for number of incontinence episodes (IEs) during Week 12 3-day diary between combination & solifenacin treatment was calculated from Mixed Effects Poisson (negative binomial) regression model including treatment group, sex, age group (<65, >=65 years), geographic region & 4-week IE reduction group as factors, log of (number of IEs/valid diary days) at baseline as covariate & log of number of valid diary days as the offset variable; Test type: Superiority; p = 0.021, Mixed Effects Poisson — p<0.05 indicates superiority in favor of treatment group with lowest rate of incontinence episodes; Rate Ratio = 0.82, 95% CI 2-sided [0.70 to 0.97], Standard Error of Mean 0.08
Statistical Analysis 4: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; EoT rate ratio, 95% CIs, & p-value for number of incontinence episodes (IEs) during EoT 3-day diary between combination & solifenacin treatment was calculated from Mixed Effects Poisson (negative binomial) regression model including treatment group, sex, age group (<65, >=65 years), geographic region & 4-week IE reduction group as factors, log of (number of IEs/valid diary days) at baseline as covariate & log of number of valid diary days as the offset variable; Test type: Superiority; p = 0.014, Mixed Effects Poisson — p<0.05 indicates superiority in favor of treatment group with lowest rate of incontinence episodes; Rate Ratio = 0.82, 95% CI 2-sided [0.71 to 0.96], Standard Error of Mean 0.08

5. Secondary Outcome: Change From Baseline in Mean Volume Voided (MVV) Per Micturition
Description: MVV per micturition was defined as MVV (mL) per micturition during last 3 days of the 3-day micturition diary period. MVV per micturition was calculated as the sum of each volume voided for each record with volume voided > 0 on valid diary days divided by the total number of records with a volume voided > 0 on valid diary days during the 3-day micturition diary period.
Time Frame: Baseline and weeks 4, 8 & 12
Population: LOCF was used for EoT. The analysis population consisted of the FAS with data available at each time point.
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Combination (Solifenacin + Mirabegron) | Solifenacin 5 mg | Solifenacin 10 mg
Number analyzed (Participants) | 707 | 705 | 698
mL
  Week 4: number analyzed (Participants) | 665 | 669 | 664
  Week 4 | 15.06 (1.55) | 11.20 (1.55) | 14.99 (1.55)
  Week 8: number analyzed (Participants) | 638 | 648 | 655
  Week 8 | 25.21 (1.89) | 14.02 (1.87) | 21.08 (1.86)
  Week 12: number analyzed (Participants) | 627 | 617 | 642
  Week 12 | 29.54 (2.06) | 17.16 (2.08) | 20.99 (2.04)
  EoT: number analyzed (Participants) | 680 | 682 | 682
  EoT | 28.05 (1.97) | 16.52 (1.97) | 20.30 (1.97)
Statistical Analysis 1: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.078, ANCOVA — P-values for pairwise comparisons were from the ANCOVA model described above. p<0.05 indicates superiority in favor of treatment group with the largest improvement; LS Means = 3.86, 95% CI 2-sided [-0.43 to 8.16], Standard Error of Mean 2.19
Statistical Analysis 2: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Means = 11.19, 95% CI 2-sided [5.98 to 16.40], Standard Error of Mean 2.66
Statistical Analysis 3: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Means = 12.38, 95% CI 2-sided [6.65 to 18.12], Standard Error of Mean 2.92
Statistical Analysis 4: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Means = 11.52, 95% CI 2-sided [6.06 to 16.99], Standard Error of Mean 2.79

6. Secondary Outcome: Change From Baseline to EoT in Corrected Micturition Frequency (CMF)
Description: CMF was defined as the mean number of micturitions per 24 hours that participants would have at EoT if their fluid intake had remained unchanged since baseline. This was calculated by the MVV per Micturition at baseline multiplied by the mean number of micturitions per 24 hours at baseline divided by the MVV per micturition at EoT.
Time Frame: Baseline and EoT (up to 12 weeks)
Population: LOCF was used. The analysis population consisted of the FAS.
Measure: Least Squares Mean (Standard Error); unit: micturitions
Arm/Group | Combination (Solifenacin + Mirabegron) | Solifenacin 5 mg | Solifenacin 10 mg
Number analyzed (Participants) | 706 | 704 | 697
micturitions | -0.96 (0.10) | -0.52 (0.10) | -0.71 (0.10)
Statistical Analysis 1: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; Adjusted change from baseline values as well as 95% CIs and p-value were generated from an ANCOVA model with treatment group, sex, age group (<65, >=65 years), 4-week incontinence reduction group and geographic region as fixed factors and baseline value as a covariate. Differences of adjusted means were calculated by subtracting adjusted mean of solifenacin monotherapy groups from adjusted mean of combination group; Test type: Superiority; p = 0.003, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Means = -0.44, 95% CI 2-sided [-0.73 to -0.16], Standard Error of Mean 0.15

7. Secondary Outcome: Change From Baseline in Mean Number of Urgency Incontinence (UI) Episodes Per 24 Hours
Description: UI was defined as the complaint of involuntary urine leakage accompanied by or immediately preceded by urgency. UI was measured using the Patient Perception of Intensity of Urgency Scale (PPIUS), a patient reported outcome validated 5-point categorical scale rating the degree of associated urinary urgency severity (0=No urgency, I felt no need to empty my bladder, but did so for other reasons. 1=Mild, I could postpone voiding as long as necessary, without fear of wetting myself. 2= Moderate, I could postpone voiding for a short while, without fear of wetting myself. 3=Severe, I could not postpone voiding, but had to rush to the toilet in order not to wet myself. 4=Urgency incontinence, I leaked before arriving to the toilet). One urgency incontinence episode was counted for each record of the diary in which the following occurred: incontinence episode or 'both' was recorded & severity of urinary urgency recorded was 3 or 4.
Time Frame: Baseline and weeks 4, 8 & 12
Population: LOCF was used for EoT. The analysis population consisted of the FAS with data available at each time point. Only participants with at least one UI episode reported in baseline diary were included.
Measure: Least Squares Mean (Standard Error); unit: UI episodes
Arm/Group | Combination (Solifenacin + Mirabegron) | Solifenacin 5 mg | Solifenacin 10 mg
Number analyzed (Participants) | 707 | 705 | 698
UI episodes
  Week 4: number analyzed (Participants) | 676 | 670 | 650
  Week 4 | -1.26 (0.07) | -0.91 (0.07) | -1.14 (0.07)
  Week 8: number analyzed (Participants) | 649 | 654 | 645
  Week 8 | -1.70 (0.07) | -1.25 (0.07) | -1.45 (0.07)
  Week 12: number analyzed (Participants) | 643 | 627 | 635
  Week 12 | -1.84 (0.07) | -1.58 (0.07) | -1.62 (0.07)
  EoT | -1.82 (0.07) | -1.54 (0.07) | -1.63 (0.07)
Statistical Analysis 1: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; Week 4 adjusted change from baseline values as well as 95% CIs were generated from an ANCOVA model with treatment group, sex, age group (<65, >=65 years), 4-week incontinence reduction group and geographic region as fixed factors and baseline value as a covariate. Differences of adjusted means were calculated by subtracting adjusted mean of solifenacin monotherapy groups from adjusted mean of combination group; Test type: Superiority; p < 0.001, stratified rank ANCOVA — P-values for pairwise comparisons were from stratified rank ANCOVA model. p<0.05 indicates superiority in favor of treatment group with the largest improvement; LS Means = -0.35, 95% CI 2-sided [-0.54 to -0.17], Standard Error of Mean 0.09
Statistical Analysis 2: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; Week 8 djusted change from baseline values as well as 95% CIs were generated from an ANCOVA model with treatment group, sex, age group (<65, >=65 years), 4-week incontinence reduction group and geographic region as fixed factors and baseline value as a covariate. Differences of adjusted means were calculated by subtracting adjusted mean of solifenacin monotherapy groups from adjusted mean of combination group; Test type: Superiority; p < 0.001, stratified rank ANCOVA — [p-value comment as in outcome 7, analysis 1]; LS Means = -0.45, 95% CI 2-sided [-0.65 to -0.25], Standard Error of Mean 0.10
Statistical Analysis 3: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; Week 12 adjusted change from baseline values as well as 95% CIs were generated from an ANCOVA model with treatment group, sex, age group (<65, >=65 years), 4-week incontinence reduction group and geographic region as fixed factors and baseline value as a covariate. Differences of adjusted means were calculated by subtracting adjusted mean of solifenacin monotherapy groups from adjusted mean of combination group; Test type: Superiority; p = 0.004, stratified rank ANCOVA — [p-value comment as in outcome 7, analysis 1]; LS Means = -0.26, 95% CI 2-sided [-0.47 to -0.05], Standard Error of Mean 0.11
Statistical Analysis 4: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; EoT adjusted change from baseline values as well as 95% CIs were generated from an ANCOVA model with treatment group, sex, age group (<65, >=65 years), 4-week incontinence reduction group and geographic region as fixed factors and baseline value as a covariate. Differences of adjusted means were calculated by subtracting adjusted mean of solifenacin monotherapy groups from adjusted mean of combination group; Test type: Superiority; p = 0.003, stratified rank ANCOVA — [p-value comment as in outcome 7, analysis 1]; LS Means = -0.27, 95% CI 2-sided [-0.47 to -0.07], Standard Error of Mean 0.10

8. Secondary Outcome: Number of UI Episodes Reported During the 3-Day Diary
Description: Number of UI episodes was calculated using the number of UI episodes recorded on valid diary days during the 3-day micturition diary period. NOTE: Only urgency incontinence episodes recorded on a valid diary day were counted.
Time Frame: Weeks 4, 8 and 12
Population: as for outcome 7
Measure: Mean (Standard Error); unit: UI episodes
Arm/Group | Combination (Solifenacin + Mirabegron) | Solifenacin 5 mg | Solifenacin 10 mg
Number analyzed (Participants) | 707 | 705 | 698
UI episodes
  Week 4: number analyzed (Participants) | 676 | 670 | 650
  Week 4 | 4.96 (0.27) | 5.86 (0.29) | 5.50 (0.30)
  Week 8: number analyzed (Participants) | 649 | 654 | 645
  Week 8 | 3.55 (0.25) | 4.76 (0.27) | 4.50 (0.30)
  Week 12: number analyzed (Participants) | 643 | 627 | 635
  Week 12 | 3.10 (0.24) | 3.78 (0.25) | 3.91 (0.30)
  EoT: number analyzed (Participants) | 691 | 683 | 666
  EoT | 3.33 (0.24) | 4.00 (0.25) | 3.96 (0.29)
Statistical Analysis 1: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; Week 4 rate ratio, 95% CIs, and p-value for number of UI episodes during Week 4 3-day diary between combination and solifenacin treatment was calculated from a Mixed Effects Poisson (negative binomial) regression model including treatment group, sex, age group (<65, >=65 years), geographic region and 4-week incontinence episode reduction group as factors, log of (number of UI episodes/number of valid diary days) at baseline as covariate and log of number of valid diary as the offset variable; Test type: Superiority; p = 0.003, Mixed Effects Poisson — p<0.05 indicates superiority in favor of treatment group with lowest rate of UI episodes; Rate Ratio = 0.85, 95% CI 2-sided [0.76 to 0.94], Standard Error of Mean 0.05
Statistical Analysis 2: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; Week 8 rate ratio, 95% CIs, and p-value for number of UI episodes during Week 8 3-day diary between combination and solifenacin treatment was calculated from a Mixed Effects Poisson (negative binomial) regression model including treatment group, sex, age group (<65, >=65 years), geographic region and 4-week incontinence episode reduction group as factors, log of (number of UI episodes/number of valid diary days) at baseline as covariate and log of number of valid diary as the offset variable; Test type: Superiority; p < 0.001, Mixed Effects Poisson — p<0.05 indicates superiority in favor of treatment group with lowest rate of UI episodes; Rate Ratio = 0.74, 95% CI 2-sided [0.63 to 0.86], Standard Error of Mean 0.08
Statistical Analysis 3: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; Week 12 rate ratio, 95% CIs, and p-value for number of UI episodes during Week 12 3-day diary between combination and solifenacin treatment was calculated from a Mixed Effects Poisson (negative binomial) regression model including treatment group, sex, age group (<65, >=65 years), geographic region and 4-week incontinence episode reduction group as factors, log of (number of UI episodes/number of valid diary days) at baseline as covariate and log of number of valid diary as the offset variable; Test type: Superiority; p = 0.038, Mixed Effects Poisson — p<0.05 indicates superiority in favor of treatment group with lowest rate of UI episodes; Rate Ratio = 0.83, 95% CI 2-sided [0.69 to 0.99], Standard Error of Mean 0.09
Statistical Analysis 4: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; EoT rate ratio, 95% CIs, and p-value for number of UI episodes during EoT 3-day diary between combination and solifenacin treatment was calculated from a Mixed Effects Poisson (negative binomial) regression model including treatment group, sex, age group (<65, >=65 years), geographic region and 4-week incontinence episode reduction group as factors, log of (number of UI episodes/number of valid diary days) at baseline as covariate and log of number of valid diary as the offset variable; Test type: Superiority; p = 0.022, Mixed Effects Poisson — p<0.05 indicates superiority in favor of treatment group with lowest rate of UI episodes; Rate Ratio = 0.82, 95% CI 2-sided [0.69 to 0.97], Standard Error of Mean 0.09

9. Secondary Outcome: Change From Baseline in Mean Number of Urgency Episodes (Grade 3 and/or 4) Per 24 Hours
Description: An urgency episode was defined as the complaint of a sudden, compelling desire to pass urine, which is difficult to defer. The mean number of urgency episodes (severity of 3 or 4) per 24 hours was defined as the average number of times a participant recorded an urgency episode (severity of 3 or 4) with or without incontinence per day during the 3-day micturition diary period. Measured using the PPIUS scale. This was calculated using the sum of each record with an urgency episode (severity of 3 or 4) recorded on a valid diary day divided by the number of valid diary days during the 3-day micturition diary period.
Time Frame: Baseline and weeks 4, 8 & 12
Population: LOCF was used for EoT. The analysis population consisted of the FAS with data available at each time point. Only participants with at least one urgency episode reported in baseline diary were included.
Measure: Least Squares Mean (Standard Error); unit: urgency episodes
Arm/Group | Combination (Solifenacin + Mirabegron) | Solifenacin 5 mg | Solifenacin 10 mg
Number analyzed (Participants) | 707 | 705 | 698
urgency episodes
  Week 4: number analyzed (Participants) | 684 | 681 | 663
  Week 4 | -1.84 (0.09) | -1.39 (0.09) | -1.74 (0.10)
  Week 8: number analyzed (Participants) | 654 | 665 | 659
  Week 8 | -2.64 (0.10) | -2.00 (0.10) | -2.29 (0.10)
  Week 12: number analyzed (Participants) | 647 | 638 | 648
  Week 12 | -2.97 (0.11) | -2.44 (0.11) | -2.55 (0.11)
  EoT: number analyzed (Participants) | 699 | 694 | 680
  EoT | -2.95 (0.10) | -2.41 (0.10) | -2.54 (0.11)
Statistical Analysis 1: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.001, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Means = -0.45, 95% CI 2-sided [-0.72 to -0.19], Standard Error of Mean 0.13
Statistical Analysis 2: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; Week 8 adjusted change from baseline values as well as 95% CIs were generated from an ANCOVA model with treatment group, sex, age group (<65, >=65 years), 4-week incontinence reduction group and geographic region as fixed factors and baseline value as a covariate. Differences of adjusted means were calculated by subtracting adjusted mean of solifenacin monotherapy groups from adjusted mean of combination group; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Means = -0.64, 95% CI 2-sided [-0.93 to -0.35], Standard Error of Mean 0.15
Statistical Analysis 3: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 7, analysis 3]; Test type: Superiority; p = 0.001, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Means = -0.52, 95% CI 2-sided [-0.82 to -0.22], Standard Error of Mean 0.15
Statistical Analysis 4: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 7, analysis 4]; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Means = -0.54, 95% CI 2-sided [-0.83 to -0.25], Standard Error of Mean 0.15

10. Secondary Outcome: Change From Baseline in Mean Number of Pads Per 24 Hours
Description: The mean number of pads per 24 hours was defined as the average number of times a participant recorded a new pad used per day during the 3-day micturition diary period. This was calculated using the number of new pads used during valid diary days during the 3-day micturition diary period divided by the number of valid diary days during the 3-day micturition diary period.
Time Frame: Baseline and weeks 4, 8 & 12
Population: LOCF was used for EoT. The analysis population consisted of the FAS with data available at each time point. Only participants with reported use of at least one pad reported in baseline diary were included.
Measure: Least Squares Mean (Standard Error); unit: pads
Arm/Group | Combination (Solifenacin + Mirabegron) | Solifenacin 5 mg | Solifenacin 10 mg
Number analyzed (Participants) | 707 | 705 | 698
pads
  Week 4: number analyzed (Participants) | 497 | 467 | 474
  Week 4 | -1.12 (0.07) | -0.86 (0.07) | -1.04 (0.07)
  Week 8: number analyzed (Participants) | 482 | 459 | 469
  Week 8 | -1.50 (0.07) | -1.17 (0.08) | -1.36 (0.08)
  Week 12: number analyzed (Participants) | 477 | 440 | 468
  Week 12 | -1.65 (0.07) | -1.38 (0.07) | -1.43 (0.07)
  EoT: number analyzed (Participants) | 510 | 476 | 487
  EoT | -1.66 (0.07) | -1.35 (0.07) | -1.43 (0.07)
Statistical Analysis 1: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; Week 4 adjusted change from baseline values as well as 95% CIs were generated from an ANCOVA model with treatment group, sex, age group (<65, >=65 years), 4-week incontinence reduction group & geographic region as fixed factors and baseline value as a covariate. Differences of adjusted means were calculated by subtracting adjusted mean of solifenacin monotherapy groups from adjusted mean of combination group; Test type: Superiority; p = 0.008, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Means = -0.26, 95% CI 2-sided [-0.46 to -0.07], Standard Error of Mean 0.10
Statistical Analysis 2: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; Week 8 adjusted change from baseline values as well as 95% CIs were generated from an ANCOVA model with treatment group, sex, age group (<65, >=65 years), 4-week incontinence reduction group & geographic region as fixed factors and baseline value as a covariate. Differences of adjusted means were calculated by subtracting adjusted mean of solifenacin monotherapy groups from adjusted mean of combination group; Test type: Superiority; p = 0.002, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Means = -0.34, 95% CI 2-sided [-0.55 to -0.13], Standard Error of Mean 0.11
Statistical Analysis 3: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; Week 12 adjusted change from baseline values as well as 95% CIs were generated from an ANCOVA model with treatment group, sex, age group (<65, >=65 years), 4-week incontinence reduction group & geographic region as fixed factors and baseline value as a covariate. Differences of adjusted means were calculated by subtracting adjusted mean of solifenacin monotherapy groups from adjusted mean of combination group; Test type: Superiority; p = 0.006, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Means = -0.28, 95% CI 2-sided [-0.47 to -0.08], Standard Error of Mean 0.10
Statistical Analysis 4: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; EoT adjusted change from baseline values as well as 95% CIs were generated from an ANCOVA model with treatment group, sex, age group (<65, >=65 years), 4-week incontinence reduction group & geographic region as fixed factors and baseline value as a covariate. Differences of adjusted means were calculated by subtracting adjusted mean of solifenacin monotherapy groups from adjusted mean of combination group; Test type: Superiority; p = 0.002, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Means = -0.31, 95% CI 2-sided [-0.51 to -0.12], Standard Error of Mean 0.10

11. Secondary Outcome: Number of Pads Used During the 3-Day Diary
Description: The number of pads used was defined as the number of times a participant recorded a new pad used during the 3-day micturition diary period. This was calculated using the sum of each record with new pad checked. Only records with new pad checked on a valid diary day were counted.
Time Frame: Weeks 4, 8 and 12
Population: LOCF was used for EoT. The analysis population consisted of the FAS with data available at each time point. Only participants who reported use of at least one pad in baseline diary were included.
Measure: Mean (Standard Error); unit: pads
Arm/Group | Combination (Solifenacin + Mirabegron) | Solifenacin 5 mg | Solifenacin 10 mg
Number analyzed (Participants) | 707 | 705 | 698
pads
  Week 4: number analyzed (Participants) | 497 | 467 | 474
  Week 4 | 4.80 (0.28) | 5.69 (0.36) | 5.41 (0.29)
  Week 8: number analyzed (Participants) | 482 | 459 | 469
  Week 8 | 3.64 (0.24) | 4.71 (0.37) | 4.50 (0.29)
  Week 12: number analyzed (Participants) | 477 | 440 | 468
  Week 12 | 3.23 (0.22) | 4.13 (0.28) | 4.07 (0.28)
  EoT: number analyzed (Participants) | 510 | 476 | 487
  EoT | 3.29 (0.22) | 4.27 (0.28) | 4.17 (0.29)
Statistical Analysis 1: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; Week 4 rate ratio, 95% CIs, and p-value for number of pads used during the 3-day diary between combination & solifenacin treatment was calculated from a Mixed Effects Poisson (negative binomial) regression model including treatment group, sex, age group (<65, >=65 years), geographic region and 4-week incontinence episode reduction group as factors, log of (number of pads used/number of valid diary days) at baseline as covariate and log of number of valid diary days as the offset variable; Test type: Superiority; p = 0.545, Mixed Effects Poisson — p<0.05 indicates superiority in favor of treatment group with lowest rate of pads used; Rate Ratio = 0.97, 95% CI 2-sided [0.87 to 1.08], Standard Error of Mean 0.06
Statistical Analysis 2: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; Week 8 rate ratio, 95% CIs, and p-value for number of pads used during the 3-day diary between combination & solifenacin treatment was calculated from a Mixed Effects Poisson (negative binomial) regression model including treatment group, sex, age group (<65, >=65 years), geographic region and 4-week incontinence episode reduction group as factors, log of (number of pads used/number of valid diary days) at baseline as covariate and log of number of valid diary days as the offset variable; Test type: Superiority; p = 0.010, Mixed Effects Poisson — p<0.05 indicates superiority in favor of treatment group with lowest rate of pads used; Rate Ratio = 0.82, 95% CI 2-sided [0.70 to 0.95], Standard Error of Mean 0.08
Statistical Analysis 3: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; Week 12 rate ratio, 95% CIs, and p-value for number of pads used during the 3-day diary between combination & solifenacin treatment was calculated from a Mixed Effects Poisson (negative binomial) regression model including treatment group, sex, age group (<65, >=65 years), geographic region and 4-week incontinence episode reduction group as factors, log of (number of pads used/number of valid diary days) at baseline as covariate and log of number of valid diary days as the offset variable; Test type: Superiority; p = 0.007, Mixed Effects Poisson — p<0.05 indicates superiority in favor of treatment group with lowest rate of pads used; Rate Ratio = 0.79, 95% CI 2-sided [0.67 to 0.94], Standard Error of Mean 0.09
Statistical Analysis 4: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; EoT rate ratio, 95% CIs, and p-value for number of pads used during the 3-day diary between combination & solifenacin treatment was calculated from a Mixed Effects Poisson (negative binomial) regression model including treatment group, sex, age group (<65, >=65 years), geographic region and 4-week incontinence episode reduction group as factors, log of (number of pads used/number of valid diary days) at baseline as covariate and log of number of valid diary days as the offset variable; Test type: Superiority; p = 0.003, Mixed Effects Poisson — p<0.05 indicates superiority in favor of treatment group with lowest rate of pads used; Rate Ratio = 0.78, 95% CI 2-sided [0.66 to 0.92], Standard Error of Mean 0.08

12. Secondary Outcome: Change From Baseline in Mean Number of Nocturia Episodes
Description: Mean number of nocturia episodes was defined as the number of times a participant urinated (excluding incontinence only episodes) while sleeping during the 3-day diary period, divided by the number of valid diary days during the diary period. Night time episode of incontinence only was not considered a nocturia episode. Nocturia episodes were counted for each micturition record which occurred between the date/time of going to bed with intention to sleep and the date/time of getting up with intention to stay awake on a valid diary day & which was accompanied by a sleep interruption. Nocturia only determined for those who were not night-shift workers.
Time Frame: Baseline and weeks 4, 8 & 12
Population: LOCF was used for EoT. The analysis population consisted of the FAS with data available at each time point. Only participants with at least one nocturia episode reported in baseline diary were included.
Measure: Least Squares Mean (Standard Error); unit: nocturia episodes
Arm/Group | Combination (Solifenacin + Mirabegron) | Solifenacin 5 mg | Solifenacin 10 mg
Number analyzed (Participants) | 707 | 705 | 698
nocturia episodes
  Week 4: number analyzed (Participants) | 526 | 514 | 517
  Week 4 | -0.28 (0.03) | -0.27 (0.03) | -0.29 (0.03)
  Week 8: number analyzed (Participants) | 500 | 501 | 514
  Week 8 | -0.37 (0.03) | -0.35 (0.03) | -0.37 (0.03)
  Week 12: number analyzed (Participants) | 492 | 480 | 510
  Week 12 | -0.46 (0.03) | -0.38 (0.03) | -0.41 (0.03)
  EoT: number analyzed (Participants) | 537 | 523 | 531
  EoT | -0.43 (0.03) | -0.37 (0.03) | -0.41 (0.03)
Statistical Analysis 1: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.836, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Means = -0.01, 95% CI 2-sided [-0.10 to 0.08], Standard Error of Mean 0.05
Statistical Analysis 2: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.617, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Means = -0.02, 95% CI 2-sided [-0.12 to 0.07], Standard Error of Mean 0.05
Statistical Analysis 3: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.134, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Means = -0.07, 95% CI 2-sided [-0.17 to 0.02], Standard Error of Mean 0.05
Statistical Analysis 4: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.174, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Means = -0.06, 95% CI 2-sided [-0.16 to 0.03], Standard Error of Mean 0.05

13. Secondary Outcome: Number of Nocturia Episodes Reported Over 3-Day Diary
Description: The number of nocturia episodes was defined as the number of times a participant urinated (excluding incontinence only episodes) during sleeping time during the 3-day micturition diary period. This was calculated using the sum of each nocturia episode recorded on valid diary days during the 3-day micturition diary period.
Time Frame: Weeks 4, 8 and 12
Population: as for outcome 12
Measure: Mean (Standard Error); unit: nocturia episodes
Arm/Group | Combination (Solifenacin + Mirabegron) | Solifenacin 5 mg | Solifenacin 10 mg
Number analyzed (Participants) | 707 | 705 | 698
nocturia episodes
  Week 4: number analyzed (Participants) | 526 | 514 | 517
  Week 4 | 3.63 (0.12) | 3.59 (0.12) | 3.58 (0.12)
  Week 8: number analyzed (Participants) | 500 | 501 | 514
  Week 8 | 3.33 (0.12) | 3.35 (0.12) | 3.32 (0.12)
  Week 12: number analyzed (Participants) | 492 | 480 | 510
  Week 12 | 3.12 (0.13) | 3.26 (0.12) | 3.23 (0.12)
  EoT: number analyzed (Participants) | 537 | 523 | 531
  EoT | 3.16 (0.12) | 3.28 (0.11) | 3.19 (0.12)
Statistical Analysis 1: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; Week 4 rate ratio, 95% CIs, & p-value for number of nocturia episodes during 3-day diary between combination & solifenacin treatment calculated from a Mixed Effects Poisson (negative binomial) regression model including treatment group, sex, age group (<65, >=65 years), geographic region & 4-week incontinence episode reduction group as factors, log of (number of nocturia episodes/number of valid diary days) at baseline as covariate and log of number of valid diary days as the offset variable; Test type: Superiority; p = 0.993, Mixed Effects Poisson — p<0.05 indicates superiority in favor of treatment group with lowest rate of nocturia episodes; Rate Ratio = 1.00, 95% CI 2-sided [0.93 to 1.08], Standard Error of Mean 0.04
Statistical Analysis 2: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; Week 8 rate ratio, 95% CIs, & p-value for number of nocturia episodes during 3-day diary between combination & solifenacin treatment calculated from a Mixed Effects Poisson (negative binomial) regression model including treatment group, sex, age group (<65, >=65 years), geographic region & 4-week incontinence episode reduction group as factors, log of (number of nocturia episodes/number of valid diary days) at baseline as covariate and log of number of valid diary days as the offset variable; Test type: Superiority; p = 0.736, Mixed Effects Poisson — p<0.05 indicates superiority in favor of treatment group with lowest rate of nocturia episodes; Rate Ratio = 0.99, 95% CI 2-sided [0.90 to 1.07], Standard Error of Mean 0.04
Statistical Analysis 3: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; Week 12 rate ratio, 95% CIs, & p-value for number of nocturia episodes during 3-day diary between combination & solifenacin treatment calculated from a Mixed Effects Poisson (negative binomial) regression model including treatment group, sex, age group (<65, >=65 years), geographic region & 4-week incontinence episode reduction group as factors, log of (number of nocturia episodes/number of valid diary days) at baseline as covariate and log of number of valid diary days as the offset variable; Test type: Superiority; p = 0.121, Mixed Effects Poisson — p<0.05 indicates superiority in favor of treatment group with lowest rate of nocturia episodes; Rate Ratio = 0.93, 95% CI 2-sided [0.85 to 1.02], Standard Error of Mean 0.05
Statistical Analysis 4: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; EoT rate ratio, 95% CIs, & p-value for number of nocturia episodes during 3-day diary between combination & solifenacin treatment calculated from a Mixed Effects Poisson (negative binomial) regression model including treatment group, sex, age group (<65, >=65 years), geographic region & 4-week incontinence episode reduction group as factors, log of (number of nocturia episodes/number of valid diary days) at baseline as covariate and log of number of valid diary days as the offset variable; Test type: Superiority; p = 0.172, Mixed Effects Poisson — p<0.05 indicates superiority in favor of treatment group with lowest rate of nocturia episodes; Rate Ratio = 0.94, 95% CI 2-sided [0.86 to 1.03], Standard Error of Mean 0.04

14. Secondary Outcome: Number of Participants With Change From Baseline to EoT in Euroqol European Quality of Life-5 Dimensions (EQ-5D) Subscale Score: Mobility
Description: The EQ-5D is an international, standardized, nondisease specific instrument for describing and valuing health status. It has 5 dimensions: Mobility, Self-care, Usual Activities, Pain/Discomfort, and Anxiety/Depression. Each dimension has 5 response levels: level 1=no problem or none; level 2=slight problems; level 3=moderate problems; level 4=severe problems; level 5=unable to perform activity.
Time Frame: Baseline and EoT (up to 12 weeks)
Population: LOCF was used for EoT. The analysis population consisted of the FAS.
Measure: Number; unit: participants
Arm/Group | Combination (Solifenacin + Mirabegron) | Solifenacin 5 mg | Solifenacin 10 mg
Number analyzed (Participants) | 707 | 705 | 698
participants
  No problems -> no problems | 409 | 370 | 374
  No problems -> slight problems | 33 | 35 | 36
  No problems -> moderate problems | 14 | 11 | 11
  No problems -> severe problems | 0 | 7 | 4
  No problems -> extreme problems | 0 | 1 | 0
  No problems -> no data | 2 | 4 | 5
  Slight problems -> no problems | 52 | 58 | 60
  Slight problems -> slight problems | 43 | 46 | 40
  Slight problems -> moderate problems | 15 | 28 | 16
  Slight problems -> severe problems | 1 | 3 | 3
  Slight problems -> extreme problems | 0 | 0 | 0
  Slight problems -> no data | 2 | 0 | 0
  Moderate problems -> no problems | 24 | 36 | 25
  Moderate problems -> slight problems | 25 | 18 | 23
  Moderate problems -> moderate problems | 28 | 28 | 40
  Moderate problems -> severe problems | 2 | 3 | 7
  Moderate problems -> extreme problems | 0 | 1 | 0
  Moderate problems -> no data | 1 | 0 | 0
  Severe problems -> no problems | 7 | 8 | 2
  Severe problems -> slight problems | 6 | 7 | 7
  Severe problems -> moderate problems | 17 | 11 | 11
  Severe problems -> severe problems | 12 | 10 | 14
  Severe problems -> extreme problems | 0 | 0 | 0
  Severe problems -> no data | 1 | 1 | 0
  Extreme problems -> no problems | 3 | 2 | 2
  Extreme problems -> slight problems | 1 | 0 | 0
  Extreme problems -> moderate problems | 1 | 1 | 1
  Extreme problems -> severe problems | 1 | 0 | 0
  Extreme problems -> extreme problems | 0 | 0 | 0
  Extreme problems -> no data | 0 | 0 | 0
  No data -> no problems | 4 | 9 | 13
  No data -> slight problems | 2 | 4 | 1
  No data -> moderate problems | 0 | 3 | 3
  No data -> severe problems | 0 | 0 | 0
  No data -> extreme problems | 0 | 0 | 0
  No data -> no data | 1 | 0 | 0

15. Secondary Outcome: Number of Participants With Change From Baseline to EoT in EQ-5D Subscale Score: Self-care
Description: as for outcome 14
Time Frame: Baseline and EoT (up to 12 weeks)
Population: LOCF was used for EoT. The analysis population consisted of the FAS.
Measure: Number; unit: participants
Arm/Group | Combination (Solifenacin + Mirabegron) | Solifenacin 5 mg | Solifenacin 10 mg
Number analyzed (Participants) | 707 | 705 | 698
participants
  No problems -> no problems | 548 | 541 | 548
  No problems -> slight problems | 28 | 26 | 25
  No problems -> moderate problems | 0 | 14 | 7
  No problems -> severe problems | 3 | 0 | 2
  No problems -> extreme problems | 0 | 0 | 0
  No problems -> no data | 6 | 5 | 4
  Slight problems -> no problems | 37 | 25 | 32
  Slight problems -> slight problems | 23 | 24 | 22
  Slight problems -> moderate problems | 9 | 7 | 9
  Slight problems -> severe problems | 1 | 0 | 0
  Slight problems -> extreme problems | 0 | 0 | 0
  Slight problems -> no data | 0 | 0 | 1
  Moderate problems -> no problems | 12 | 16 | 7
  Moderate problems -> slight problems | 9 | 9 | 5
  Moderate problems -> moderate problems | 11 | 7 | 12
  Moderate problems -> severe problems | 0 | 2 | 2
  Moderate problems -> extreme problems | 0 | 0 | 0
  Moderate problems -> no data | 0 | 0 | 0
  Severe problems -> no problems | 7 | 5 | 0
  Severe problems -> slight problems | 2 | 2 | 2
  Severe problems -> moderate problems | 2 | 1 | 2
  Severe problems -> severe problems | 1 | 4 | 1
  Severe problems -> extreme problems | 0 | 0 | 0
  Severe problems -> no data | 0 | 0 | 0
  Extreme problems -> no problems | 0 | 0 | 0
  Extreme problems -> slight problems | 0 | 1 | 0
  Extreme problems -> moderate problems | 0 | 0 | 0
  Extreme problems -> severe problems | 1 | 0 | 0
  Extreme problems -> extreme problems | 0 | 0 | 0
  Extreme problems -> no data | 0 | 0 | 0
  No data -> no problems | 6 | 14 | 17
  No data -> slight problems | 0 | 2 | 0
  No data -> moderate problems | 0 | 0 | 0
  No data -> severe problems | 0 | 0 | 0
  No data -> extreme problems | 0 | 0 | 0
  No data -> no data | 1 | 0 | 0

16. Secondary Outcome: Number of Participants With Change From Baseline to EoT in EQ-5D Subscale Score: Usual Activities
Description: as for outcome 14
Time Frame: Baseline and EoT (up to 12 weeks)
Population: LOCF was used for EoT. The analysis population consisted of the FAS.
Measure: Number; unit: participants
Arm/Group | Combination (Solifenacin + Mirabegron) | Solifenacin 5 mg | Solifenacin 10 mg
Number analyzed (Participants) | 707 | 705 | 698
participants
  No problems -> no problems | 397 | 384 | 379
  No problems -> slight problems | 38 | 30 | 42
  No problems -> moderate problems | 12 | 19 | 11
  No problems -> severe problems | 1 | 4 | 1
  No problems -> extreme problems | 0 | 0 | 1
  No problems -> no data | 4 | 3 | 3
  Slight problems -> no problems | 75 | 81 | 78
  Slight problems -> slight problems | 46 | 45 | 37
  Slight problems -> moderate problems | 12 | 16 | 15
  Slight problems -> severe problems | 1 | 1 | 3
  Slight problems -> extreme problems | 0 | 1 | 0
  Slight problems -> no data | 0 | 1 | 2
  Moderate problems -> no problems | 29 | 35 | 25
  Moderate problems -> slight problems | 22 | 20 | 28
  Moderate problems -> moderate problems | 22 | 18 | 21
  Moderate problems -> severe problems | 3 | 3 | 4
  Moderate problems -> extreme problems | 1 | 0 | 0
  Moderate problems -> no data | 2 | 1 | 0
  Severe problems -> no problems | 9 | 8 | 12
  Severe problems -> slight problems | 7 | 5 | 1
  Severe problems -> moderate problems | 7 | 6 | 9
  Severe problems -> severe problems | 5 | 7 | 9
  Severe problems -> extreme problems | 0 | 0 | 0
  Severe problems -> no data | 0 | 0 | 0
  Extreme problems -> no problems | 2 | 0 | 0
  Extreme problems -> slight problems | 1 | 0 | 0
  Extreme problems -> moderate problems | 3 | 1 | 0
  Extreme problems -> severe problems | 1 | 0 | 0
  Extreme problems -> extreme problems | 0 | 0 | 0
  Extreme problems -> no data | 0 | 0 | 0
  No data -> no problems | 5 | 11 | 15
  No data -> slight problems | 1 | 4 | 1
  No data -> moderate problems | 0 | 1 | 1
  No data -> severe problems | 0 | 0 | 0
  No data -> extreme problems | 0 | 0 | 0
  No data -> no data | 1 | 0 | 0

17. Secondary Outcome: Number of Participants With Change From Baseline to EoT in EQ-5D Subscale Score: Pain/Discomfort
Description: as for outcome 14
Time Frame: Baseline and EoT (up to 12 weeks)
Population: LOCF was used for EoT. The analysis population consisted of the FAS.
Measure: Number; unit: participants
Arm/Group | Combination (Solifenacin + Mirabegron) | Solifenacin 5 mg | Solifenacin 10 mg
Number analyzed (Participants) | 707 | 705 | 698
participants
  No pain -> no pain | 299 | 290 | 283
  No pain -> slight pain | 45 | 62 | 51
  No pain -> moderate pain | 12 | 14 | 17
  No pain -> severe pain | 3 | 9 | 2
  No pain -> extreme pain | 0 | 0 | 1
  No pain -> no data | 4 | 4 | 3
  Slight pain -> no pain | 79 | 82 | 81
  Slight pain -> slight pain | 58 | 64 | 55
  Slight pain -> moderate pain | 28 | 17 | 31
  Slight pain -> severe pain | 0 | 2 | 5
  Slight pain -> extreme pain | 1 | 2 | 0
  Slight pain -> no data | 0 | 0 | 2
  Moderate pain -> no pain | 39 | 36 | 21
  Moderate pain -> slight pain | 37 | 36 | 39
  Moderate pain -> moderate pain | 34 | 30 | 39
  Moderate pain -> severe pain | 7 | 4 | 8
  Moderate pain -> extreme pain | 0 | 1 | 0
  Moderate pain -> no data | 2 | 1 | 0
  Severe pain -> no pain | 7 | 4 | 10
  Severe pain -> slight pain | 12 | 7 | 4
  Severe pain -> moderate pain | 11 | 16 | 16
  Severe pain -> severe pain | 10 | 4 | 9
  Severe pain -> extreme pain | 0 | 1 | 1
  Severe pain -> no data | 0 | 0 | 0
  Extreme pain -> no pain | 4 | 1 | 0
  Extreme pain -> slight pain | 0 | 1 | 1
  Extreme pain -> moderate pain | 1 | 0 | 1
  Extreme pain -> severe pain | 6 | 1 | 1
  Extreme pain -> extreme pain | 1 | 0 | 0
  Extreme pain -> no data | 0 | 0 | 0
  No data -> no pain | 4 | 8 | 11
  No data -> slight pain | 1 | 3 | 4
  No data -> moderate pain | 1 | 5 | 2
  No data -> severe pain | 0 | 0 | 0
  No data -> extreme pain | 0 | 0 | 0
  No data -> no data | 1 | 0 | 0

18. Secondary Outcome: Number of Participants With Change From Baseline to EoT in EQ-5D Subscale Score: Anxiety/Depression
Description: as for outcome 14
Time Frame: Baseline and EoT (up to 12 weeks)
Population: LOCF was used for EoT. The analysis population consisted of the FAS.
Measure: Number; unit: participants
Arm/Group | Combination (Solifenacin + Mirabegron) | Solifenacin 5 mg | Solifenacin 10 mg
Number analyzed (Participants) | 707 | 705 | 698
participants
  Not anxious -> not anxious | 322 | 300 | 307
  Not anxious -> slightly anxious | 43 | 39 | 43
  Not anxious -> moderately anxious | 11 | 17 | 15
  Not anxious -> severely anxious | 2 | 2 | 3
  Not anxious-> extremely anxious | 0 | 0 | 0
  Not anxious -> no data | 4 | 3 | 3
  Slightly anxious -> not anxious | 107 | 99 | 90
  Slightly anxious -> slightly anxious | 56 | 60 | 69
  Slightly anxious -> moderately anxious | 13 | 11 | 23
  Slightly anxious -> severely anxious | 1 | 2 | 2
  Slightly anxious -> extremely anxious | 0 | 0 | 0
  Slightly anxious -> no data | 1 | 2 | 2
  Moderately anxious -> not anxious | 36 | 38 | 34
  Moderately anxious -> slightly anxious | 36 | 40 | 33
  Moderately anxious -> moderately anxious | 22 | 26 | 17
  Moderately anxious -> severely anxious | 3 | 7 | 1
  Moderately anxious -> extremely anxious | 0 | 3 | 1
  Moderately anxious -> no data | 0 | 0 | 0
  Severely anxious -> not anxious | 10 | 8 | 8
  Severely anxious -> slightly anxious | 9 | 5 | 5
  Severely anxious -> moderately anxious | 6 | 6 | 11
  Severely anxious -> severely anxious | 5 | 8 | 7
  Severely anxious -> extremely anxious | 0 | 3 | 0
  Severely anxious -> no data | 0 | 0 | 0
  Extremely anxious -> not anxious | 1 | 4 | 1
  Extremely anxious -> slightly anxious | 2 | 1 | 1
  Extremely anxious -> moderately anxious | 4 | 2 | 3
  Extremely anxious -> severely anxious | 4 | 1 | 1
  Extremely anxious -> extremely anxious | 1 | 2 | 1
  Extremely anxious -> no data | 1 | 0 | 0
  No data -> not anxious | 5 | 13 | 11
  No data -> slightly anxious | 0 | 2 | 5
  No data -> moderately anxious | 1 | 1 | 1
  No data -> severely anxious | 0 | 0 | 0
  No data -> extremely anxious | 0 | 0 | 0
  No data -> no data | 1 | 0 | 0

19. Secondary Outcome: Change From Baseline in Overactive Bladder Symptom (OAB-q) Symptom Bother Score
Description: The OAB-q was a self-reported questionnaire comprising 33-items each rated on a 6-point Likert scale. The questionnaire consisted of an 8-item symptom bother scale and 25 health-related QoL (HRQL) items comprising 4 HRQL subscales (Coping, Concern, Sleep, and Social Interaction). Symptom Bother score ranges from 0 (least severity) to 100 (worst severity).
Time Frame: Baseline and weeks 4, 8 & 12
Population: LOCF was used for EoT. The analysis population consisted of the FAS with data available at each time point.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Combination (Solifenacin + Mirabegron) | Solifenacin 5 mg | Solifenacin 10 mg
Number analyzed (Participants) | 707 | 705 | 698
units on a scale
  Week 4: number analyzed (Participants) | 682 | 677 | 669
  Week 4 | -16.68 (0.65) | -13.79 (0.65) | -15.82 (0.65)
  Week 8: number analyzed (Participants) | 670 | 660 | 658
  Week 8 | -22.86 (0.68) | -18.36 (0.69) | -19.34 (0.69)
  Week 12: number analyzed (Participants) | 644 | 641 | 647
  Week 12 | -27.90 (0.71) | -22.31 (0.71) | -24.09 (0.71)
  EoT: number analyzed (Participants) | 694 | 683 | 676
  EoT | -26.89 (0.69) | -21.93 (0.70) | -23.59 (0.70)
Statistical Analysis 1: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; Week 4 adjusted change from baseline values as well as 95% CIs & p-value were generated from ANCOVA model with treatment group, sex, age group (<65, >=65 years), 4-week incontinence reduction group and geographic region as fixed factors & baseline value as a covariate. Differences of adjusted means were calculated by subtracting adjusted mean of solifenacin monotherapy groups from adjusted mean of combination group; Test type: Superiority; p = 0.002, ANCOVA — P-values for pairwise comparisons were from the ANCOVA model described above. p<0.05 indicated superiority in favor of treatment group with the largest improvement; LS Means = -2.89, 95% CI 2-sided [-4.68 to -1.10], Standard Error of Mean 0.91
Statistical Analysis 2: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; Week 8 adjusted change from baseline values as well as 95% CIs & p-value were generated from ANCOVA model with treatment group, sex, age group (<65, >=65 years), 4-week incontinence reduction group and geographic region as fixed factors & baseline value as a covariate. Differences of adjusted means were calculated by subtracting adjusted mean of solifenacin monotherapy groups from adjusted mean of combination group; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 19, analysis 1]; LS Means = -4.50, 95% CI 2-sided [-6.40 to -2.60], Standard Error of Mean 0.97
Statistical Analysis 3: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; Week 12 adjusted change from baseline values as well as 95% CIs & p-value were generated from ANCOVA model with treatment group, sex, age group (<65, >=65 years), 4-week incontinence reduction group and geographic region as fixed factors & baseline value as a covariate. Differences of adjusted means were calculated by subtracting adjusted mean of solifenacin monotherapy groups from adjusted mean of combination group; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 19, analysis 1]; LS Means = -5.59, 95% CI 2-sided [-7.56 to -3.62], Standard Error of Mean 1.00
Statistical Analysis 4: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; EoT adjusted change from baseline values as well as 95% CIs & p-value were generated from ANCOVA model with treatment group, sex, age group (<65, >=65 years), 4-week incontinence reduction group and geographic region as fixed factors & baseline value as a covariate. Differences of adjusted means were calculated by subtracting adjusted mean of solifenacin monotherapy groups from adjusted mean of combination group; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 19, analysis 1]; LS Means = -4.96, 95% CI 2-sided [-6.88 to -3.04], Standard Error of Mean 0.98

20. Secondary Outcome: Change From Baseline in OAB-q Health-Related Quality of Life (HRQL) Total Score
Description: The OAB-q was a self-reported questionnaire comprising 33-items each rated on a 6-point Likert scale. The questionnaire consisted of an 8-item symptom bother scale and 25 health-related QoL (HRQL) items comprising 4 HRQL subscales (Coping, Concern, Sleep, and Social Interaction). HRQL subscales (coping, concern, sleep and social) and total score range from 0 (worst quality of life) to 100 (best quality of life).
Time Frame: Baseline and weeks 4, 8 & 12
Population: LOCF was used for EoT. The analysis population consisted of the FAS with data available at each time point.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Combination (Solifenacin + Mirabegron) | Solifenacin 5 mg | Solifenacin 10 mg
Number analyzed (Participants) | 707 | 705 | 698
units on a scale
  Week 4: number analyzed (Participants) | 682 | 677 | 669
  Week 4 | 12.95 (0.59) | 11.03 (0.59) | 12.44 (0.59)
  Week 8: number analyzed (Participants) | 670 | 660 | 658
  Week 8 | 17.58 (0.63) | 15.26 (0.63) | 14.60 (0.64)
  Week 12: number analyzed (Participants) | 644 | 641 | 647
  Week 12 | 21.40 (0.66) | 17.91 (0.67) | 17.72 (0.66)
  EoT: number analyzed (Participants) | 694 | 683 | 676
  EoT | 20.78 (0.65) | 17.63 (0.65) | 17.40 (0.65)
Statistical Analysis 1: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 19, analysis 1]; Test type: Superiority; p = 0.021, ANCOVA — [p-value comment as in outcome 19, analysis 1]; LS Means = 1.92, 95% CI 2-sided [0.29 to 3.55], Standard Error of Mean 0.83
Statistical Analysis 2: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 19, analysis 2]; Test type: Superiority; p = 0.010, ANCOVA — [p-value comment as in outcome 19, analysis 1]; LS Means = 2.31, 95% CI 2-sided [0.56 to 4.06], Standard Error of Mean 0.89
Statistical Analysis 3: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 19, analysis 3]; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 19, analysis 1]; LS Means = 3.49, 95% CI 2-sided [1.65 to 5.33], Standard Error of Mean 0.94
Statistical Analysis 4: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 19, analysis 4]; Test type: Superiority; p = 0.001, ANCOVA — [p-value comment as in outcome 19, analysis 1]; LS Means = 3.15, 95% CI 2-sided [1.35 to 4.95], Standard Error of Mean 0.92

21. Secondary Outcome: Change From Baseline in OAB-q HRQL Subscale Score: Coping
Description: as for outcome 20
Time Frame: Baseline and weeks 4, 8 & 12
Population: LOCF was used for EoT. The analysis population consisted of the FAS with data available at each time point.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Combination (Solifenacin + Mirabegron) | Solifenacin 5 mg | Solifenacin 10 mg
Number analyzed (Participants) | 707 | 705 | 698
units on a scale
  Week 4: number analyzed (Participants) | 682 | 677 | 669
  Week 4 | 15.17 (0.68) | 12.27 (0.68) | 14.25 (0.68)
  Week 8: number analyzed (Participants) | 670 | 660 | 658
  Week 8 | 20.82 (0.74) | 17.47 (0.74) | 16.87 (0.74)
  Week 12: number analyzed (Participants) | 644 | 641 | 647
  Week 12 | 25.16 (0.78) | 20.45 (0.78) | 20.20 (0.78)
  EoT: number analyzed (Participants) | 694 | 683 | 676
  EoT | 24.48 (0.75) | 20.19 (0.76) | 19.90 (0.76)
Statistical Analysis 1: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 19, analysis 1]; Test type: Superiority; p = 0.003, ANCOVA — [p-value comment as in outcome 19, analysis 1]; LS Means = 2.90, 95% CI 2-sided [1.02 to 4.78], Standard Error of Mean 0.96
Statistical Analysis 2: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 19, analysis 2]; Test type: Superiority; p = 0.001, ANCOVA — [p-value comment as in outcome 19, analysis 1]; LS Means = 3.35, 95% CI 2-sided [1.29 to 5.40], Standard Error of Mean 1.05
Statistical Analysis 3: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 19, analysis 3]; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 19, analysis 1]; LS Means = 4.71, 95% CI 2-sided [2.55 to 6.87], Standard Error of Mean 1.10
Statistical Analysis 4: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 19, analysis 4]; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 19, analysis 1]; LS Means = 4.29, 95% CI 2-sided [2.20 to 6.39], Standard Error of Mean 1.07

22. Secondary Outcome: Change From Baseline in OAB-q HRQL Subscale Score: Concern
Description: as for outcome 20
Time Frame: Baseline and weeks 4, 8 & 12
Population: LOCF was used for EoT. The analysis population consisted of the FAS with data available at each time point.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Combination (Solifenacin + Mirabegron) | Solifenacin 5 mg | Solifenacin 10 mg
Number analyzed (Participants) | 707 | 705 | 698
units on a scale
  Week 4: number analyzed (Participants) | 682 | 677 | 669
  Week 4 | 13.79 (0.68) | 11.85 (0.68) | 13.82 (0.69)
  Week 8: number analyzed (Participants) | 670 | 660 | 658
  Week 8 | 18.87 (0.70) | 16.36 (0.71) | 15.88 (0.71)
  Week 12: number analyzed (Participants) | 644 | 641 | 647
  Week 12 | 22.85 (0.74) | 19.24 (0.75) | 19.67 (0.74)
  Week EoT: number analyzed (Participants) | 694 | 683 | 676
  Week EoT | 22.28 (0.72) | 19.00 (0.73) | 19.28 (0.73)
Statistical Analysis 1: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 19, analysis 1]; Test type: Superiority; p = 0.044, ANCOVA — [p-value comment as in outcome 19, analysis 1]; LS Means = 1.94, 95% CI 2-sided [0.05 to 3.83], Standard Error of Mean 0.96
Statistical Analysis 2: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 19, analysis 2]; Test type: Superiority; p = 0.012, ANCOVA — [p-value comment as in outcome 19, analysis 1]; LS Means = 2.50, 95% CI 2-sided [0.55 to 4.46], Standard Error of Mean 1.00
Statistical Analysis 3: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 19, analysis 3]; Test type: Superiority; p = 0.001, ANCOVA — [p-value comment as in outcome 19, analysis 1]; LS Means = 3.61, 95% CI 2-sided [1.54 to 5.67], Standard Error of Mean 1.05
Statistical Analysis 4: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 19, analysis 4]; Test type: Superiority; p = 0.001, ANCOVA — [p-value comment as in outcome 19, analysis 1]; LS Means = 3.28, 95% CI 2-sided [1.27 to 5.29], Standard Error of Mean 1.03

23. Secondary Outcome: Change From Baseline in OAB-q HRQL Subscale Score: Sleep
Description: as for outcome 20
Time Frame: Baseline and weeks 4, 8 & 12
Population: LOCF was used for EoT. The analysis population consisted of the FAS with data available at each time point.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Combination (Solifenacin + Mirabegron) | Solifenacin 5 mg | Solifenacin 10 mg
Number analyzed (Participants) | 707 | 705 | 698
units on a scale
  Week 4: number analyzed (Participants) | 682 | 677 | 669
  Week 4 | 11.58 (0.68) | 11.04 (0.68) | 11.16 (0.69)
  Week 8: number analyzed (Participants) | 670 | 660 | 658
  Week 8 | 16.18 (0.71) | 14.57 (0.71) | 13.72 (0.71)
  Week 12: number analyzed (Participants) | 644 | 641 | 647
  Week 12 | 20.00 (0.74) | 17.74 (0.74) | 16.84 (0.74)
  Week EoT: number analyzed (Participants) | 694 | 683 | 676
  Week EoT | 19.16 (0.72) | 17.30 (0.73) | 16.55 (0.73)
Statistical Analysis 1: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 19, analysis 1]; Test type: Superiority; p = 0.575, ANCOVA — [p-value comment as in outcome 19, analysis 1]; LS Means = 0.54, 95% CI 2-sided [-1.35 to 2.43], Standard Error of Mean 0.96
Statistical Analysis 2: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 19, analysis 2]; Test type: Superiority; p = 0.109, ANCOVA — [p-value comment as in outcome 19, analysis 1]; LS Means = 1.61, 95% CI 2-sided [-0.36 to 3.58], Standard Error of Mean 1.00
Statistical Analysis 3: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 19, analysis 3]; Test type: Superiority; p = 0.032, ANCOVA — [p-value comment as in outcome 19, analysis 1]; LS Means = 2.26, 95% CI 2-sided [0.20 to 4.32], Standard Error of Mean 1.05
Statistical Analysis 4: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 19, analysis 4]; Test type: Superiority; p = 0.069, ANCOVA — [p-value comment as in outcome 19, analysis 1]; LS Means = 1.86, 95% CI 2-sided [-0.15 to 3.87], Standard Error of Mean 1.02

24. Secondary Outcome: Change From Baseline in OAB-q HRQL Subscale Score: Social Interaction
Description: as for outcome 20
Time Frame: Baseline and weeks 4, 8 & 12
Population: LOCF was used for EoT. The analysis population consisted of the FAS with data available at each time point.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Combination (Solifenacin + Mirabegron) | Solifenacin 5 mg | Solifenacin 10 mg
Number analyzed (Participants) | 707 | 705 | 698
units on a scale
  Week 4: number analyzed (Participants) | 682 | 677 | 669
  Week 4 | 9.58 (0.59) | 7.85 (0.59) | 8.95 (0.59)
  Week 8: number analyzed (Participants) | 670 | 660 | 658
  Week 8 | 11.93 (0.60) | 10.84 (0.60) | 10.16 (0.60)
  Week 12: number analyzed (Participants) | 644 | 641 | 647
  Week 12 | 14.70 (0.61) | 12.08 (0.61) | 11.98 (0.61)
  EoT: number analyzed (Participants) | 694 | 683 | 676
  EoT | 14.39 (0.60) | 11.91 (0.60) | 11.72 (0.61)
Statistical Analysis 1: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 19, analysis 1]; Test type: Superiority; p = 0.037, ANCOVA — [p-value comment as in outcome 19, analysis 1]; LS Means = 1.73, 95% CI 2-sided [0.10 to 3.36], Standard Error of Mean 0.83
Statistical Analysis 2: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 19, analysis 2]; Test type: Superiority; p = 0.199, ANCOVA — [p-value comment as in outcome 19, analysis 1]; LS Means = 1.09, 95% CI 2-sided [-0.57 to 2.76], Standard Error of Mean 0.85
Statistical Analysis 3: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 19, analysis 3]; Test type: Superiority; p = 0.003, ANCOVA — [p-value comment as in outcome 19, analysis 1]; LS Means = 2.62, 95% CI 2-sided [0.92 to 4.31], Standard Error of Mean 0.87
Statistical Analysis 4: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 19, analysis 4]; Test type: Superiority; p = 0.004, ANCOVA — [p-value comment as in outcome 19, analysis 1]; LS Means = 2.48, 95% CI 2-sided [0.81 to 4.15], Standard Error of Mean 0.85

25. Secondary Outcome: Change From Baseline in Treatment Satisfaction - Visual Analogue Scale (TS-VAS) Score
Description: The TS-VAS rated participant satisfaction with treatment on a scale from 0 (No, not at all) to 10 (Yes, completely).
Time Frame: Baseline and weeks 4, 8 & 12
Population: LOCF was used for EoT. The analysis population consisted of the FAS with data available at each time point.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Combination (Solifenacin + Mirabegron) | Solifenacin 5 mg | Solifenacin 10 mg
Number analyzed (Participants) | 707 | 705 | 698
units on a scale
  Week 4: number analyzed (Participants) | 680 | 677 | 668
  Week 4 | 1.2 (0.1) | 0.8 (0.1) | 1.1 (0.1)
  Week 8: number analyzed (Participants) | 668 | 660 | 656
  Week 8 | 1.5 (0.1) | 1.2 (0.1) | 1.3 (0.1)
  Week 12: number analyzed (Participants) | 644 | 641 | 646
  Week 12 | 1.9 (0.1) | 1.4 (0.1) | 1.6 (0.1)
  EoT: number analyzed (Participants) | 693 | 683 | 675
  EoT | 1.8 (0.1) | 1.4 (0.1) | 1.6 (0.1)
Statistical Analysis 1: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; Week 4 adjusted change from baseline values as well as the 95% CIs and p-value were generated from an ANCOVA model with treatment group, sex, age group (<65, >=65 years), 4-week incontinence reduction group and geographic region as fixed factors and baseline value as a covariate. Differences of adjusted means were calculated by subtracting adjusted mean of solifenacin monotherapy groups from adjusted mean of combination group; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 19, analysis 1]; LS Means = 0.4, 95% CI 2-sided [0.2 to 0.6], Standard Error of Mean 0.1
Statistical Analysis 2: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; Week 8 adjusted change from baseline values as well as the 95% CIs and p-value were generated from an ANCOVA model with treatment group, sex, age group (<65, >=65 years), 4-week incontinence reduction group and geographic region as fixed factors and baseline value as a covariate. Differences of adjusted means were calculated by subtracting adjusted mean of solifenacin monotherapy groups from adjusted mean of combination group; Test type: Superiority; p = 0.019, ANCOVA — [p-value comment as in outcome 19, analysis 1]; LS Means = 0.3, 95% CI 2-sided [0.0 to 0.5], Standard Error of Mean 0.1
Statistical Analysis 3: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; Week 12 adjusted change from baseline values as well as the 95% CIs and p-value were generated from an ANCOVA model with treatment group, sex, age group (<65, >=65 years), 4-week incontinence reduction group and geographic region as fixed factors and baseline value as a covariate. Differences of adjusted means were calculated by subtracting adjusted mean of solifenacin monotherapy groups from adjusted mean of combination group; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 19, analysis 1]; LS Means = 0.5, 95% CI 2-sided [0.3 to 0.7], Standard Error of Mean 0.1
Statistical Analysis 4: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; EoT adjusted change from baseline values as well as the 95% CIs and p-value were generated from an ANCOVA model with treatment group, sex, age group (<65, >=65 years), 4-week incontinence reduction group and geographic region as fixed factors and baseline value as a covariate. Differences of adjusted means were calculated by subtracting adjusted mean of solifenacin monotherapy groups from adjusted mean of combination group; Test type: Superiority; p = 0.001, ANCOVA — [p-value comment as in outcome 19, analysis 1]; LS Means = 0.4, 95% CI 2-sided [0.2 to 0.6], Standard Error of Mean 0.1

26. Secondary Outcome: Change From Baseline in Patient Perception Bladder Control (PPBC) Score
Description: The PPBC was a validated, global assessment tool using a 6-point Likert scale on which participants rated their subjective impression of their current bladder condition. PPBC score: 1-no problem, 2- some very minor problems, 3-some minor problems, 4-moderate problems, 5-severe problems, 6-many severe problems.
Time Frame: Baseline and weeks 4, 8 & 12
Population: LOCF was used for EoT. The analysis population consisted of the FAS with data available at each time point.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Combination (Solifenacin + Mirabegron) | Solifenacin 5 mg | Solifenacin 10 mg
Number analyzed (Participants) | 707 | 705 | 698
units on a scale
  Week 4: number analyzed (Participants) | 687 | 685 | 677
  Week 4 | -0.9 (0.0) | -0.6 (0.0) | -0.7 (0.0)
  Week 8: number analyzed (Participants) | 673 | 667 | 669
  Week 8 | -1.2 (0.0) | -1.0 (0.0) | -1.0 (0.0)
  Week 12: number analyzed (Participants) | 647 | 648 | 655
  Week 12 | -1.5 (0.0) | -1.2 (0.0) | -1.3 (0.0)
  EoT: number analyzed (Participants) | 697 | 688 | 683
  EoT | -1.5 (0.0) | -1.2 (0.0) | -1.3 (0.0)
Statistical Analysis 1: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; Week 4 adjusted change from baseline values as well as the 95% CIs and p-value were generated from ANCOVA model with treatment group, sex, age group (<65, >=65 years), 4-week incontinence reduction group and geographic region as fixed factors and baseline value as a covariate. Difference of adjusted mean was calculated by subtracting adjusted mean of solifenacin monotherapy groups from adjusted mean of combination group; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 19, analysis 1]; LS Means = -0.2, 95% CI 2-sided [-0.4 to -0.1], Standard Error of Mean 0.1
Statistical Analysis 2: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; Week 8 adjusted change from baseline values as well as the 95% CIs and p-value were generated from ANCOVA model with treatment group, sex, age group (<65, >=65 years), 4-week incontinence reduction group and geographic region as fixed factors and baseline value as a covariate. Difference of adjusted mean was calculated by subtracting adjusted mean of solifenacin monotherapy groups from adjusted mean of combination group; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 19, analysis 1]; LS Means = -0.2, 95% CI 2-sided [-0.4 to -0.1], Standard Error of Mean 0.1
Statistical Analysis 3: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; Week 12 adjusted change from baseline values as well as the 95% CIs and p-value were generated from ANCOVA model with treatment group, sex, age group (<65, >=65 years), 4-week incontinence reduction group and geographic region as fixed factors and baseline value as a covariate. Difference of adjusted mean was calculated by subtracting adjusted mean of solifenacin monotherapy groups from adjusted mean of combination group; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 19, analysis 1]; LS Means = -0.3, 95% CI 2-sided [-0.4 to -0.2], Standard Error of Mean 0.1
Statistical Analysis 4: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; EoT adjusted change from baseline values as well as the 95% CIs and p-value were generated from ANCOVA model with treatment group, sex, age group (<65, >=65 years), 4-week incontinence reduction group and geographic region as fixed factors and baseline value as a covariate. Difference of adjusted mean was calculated by subtracting adjusted mean of solifenacin monotherapy groups from adjusted mean of combination group; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 19, analysis 1]; LS Means = -0.3, 95% CI 2-sided [-0.4 to -0.1], Standard Error of Mean 0.1

27. Secondary Outcome: Number of Participants in Each Category of Patient and Clinician Global Impression of Change Scales (PGIC and CGIC)
Description: The PGIC was a 2-part questionnaire, assessing both the change in the participant's overall condition (Patient Impression in General Health (PIBS)) and change in bladder condition since the start of the study (Patient Impression in General Health (PIGH)) (from very much worse to very much improved). The CGIC was a single questionnaire assessing the participant's change in bladder condition since the beginning of the study (Clinician Impression in Bladder Symptoms (CIBS)).
Time Frame: End of treatment (up to 12 weeks)
Population: LOCF was used for EoT. The analysis population consisted of the FAS.
Measure: Number; unit: participants
Arm/Group | Combination (Solifenacin + Mirabegron) | Solifenacin 5 mg | Solifenacin 10 mg
Number analyzed (Participants) | 707 | 705 | 698
participants
  PIBS Very Much Improved | 227 | 152 | 171
  PIBS Much Improved | 257 | 264 | 284
  PIBS Minimally Improved | 135 | 170 | 152
  PIBS No Change | 25 | 55 | 56
  PIBS Minimally Worse | 7 | 11 | 4
  PIBS Much Worse | 4 | 4 | 6
  PIBS Very Much Worse | 0 | 1 | 1
  PIGH Very Much Improved | 144 | 104 | 108
  PIGH Much Improved | 239 | 236 | 244
  PIGH Minimally Improved | 143 | 147 | 146
  PIGH No Change | 113 | 142 | 160
  PIGH Minimally Worse | 14 | 23 | 10
  PIGH Much Worse | 1 | 4 | 4
  PIGH Very Much Worse | 1 | 1 | 2
  CIBS Very Much Improved | 184 | 118 | 141
  CIBS Much Improved | 311 | 316 | 329
  CIBS Minimally Improved | 141 | 164 | 155
  CIBS No Change | 23 | 56 | 40
  CIBS Minimally Worse | 4 | 8 | 5
  CIBS Much Worse | 4 | 3 | 5
  CIBS Very Much Worse | 3 | 3 | 4

28. Secondary Outcome: Percentage of Participants With at Least a 50% Decrease From Baseline in Mean Number of Incontinence Episodes Per 24 Hours
Description: Incontinence was defined as any involuntary leakage of urine.
Time Frame: Weeks 4, 8 and 12
Population: LOCF was used for EoT. The analysis population consisted of the FAS with data available at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Combination (Solifenacin + Mirabegron) | Solifenacin 5 mg | Solifenacin 10 mg
Number analyzed (Participants) | 707 | 705 | 698
percentage of participants
  Week 4: number analyzed (Participants) | 690 | 690 | 679
  Week 4 | 52.5 | 43.3 | 49.0
  Week 8: number analyzed (Participants) | 661 | 674 | 673
  Week 8 | 66.9 | 57.6 | 61.8
  Week 12: number analyzed (Participants) | 653 | 645 | 664
  Week 12 | 72.4 | 64.0 | 66.9
  EoT: number analyzed (Participants) | 706 | 704 | 697
  EoT | 71.2 | 63.1 | 66.6
Statistical Analysis 1: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; Week 4 odds ratios, 95% Two sided CIs for Odds ratios and p-values were from a logistic regression model including treatment group, sex, age group (<65, >=65 years), 4-week incontinence episode reduction group, geographic region as factors and baseline value as covariate; Test type: Superiority; p < 0.001, Regression, Logistic — p<0.05 indicated superiority in favor of treatment group with highest response; Odds Ratio (OR) = 1.48, 95% CI 2-sided [1.19 to 1.84]
Statistical Analysis 2: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; Week 8 odds ratios, 95% Two sided CIs for Odds ratios and p-values were from a logistic regression model including treatment group, sex, age group (<65, >=65 years), 4-week incontinence episode reduction group, geographic region as factors and baseline value as covariate; Test type: Superiority; p < 0.001, Regression, Logistic — p<0.05 indicated superiority in favor of treatment group with highest response; Odds Ratio (OR) = 1.57, 95% CI 2-sided [1.25 to 1.98]
Statistical Analysis 3: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; Week 12 odds ratios, 95% Two sided CIs for Odds ratios and p-values were from a logistic regression model including treatment group, sex, age group (<65, >=65 years), 4-week incontinence episode reduction group, geographic region as factors and baseline value as covariate; Test type: Superiority; p = 0.001, Regression, Logistic — p<0.05 indicated superiority in favor of treatment group with highest response; Odds Ratio (OR) = 1.54, 95% CI 2-sided [1.21 to 1.95]
Statistical Analysis 4: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; EoT odds ratios, 95% Two sided CIs for Odds ratios and p-values were from a logistic regression model including treatment group, sex, age group (<65, >=65 years), 4-week incontinence episode reduction group, geographic region as factors and baseline value as covariate; Test type: Superiority; p < 0.001, Regression, Logistic — p<0.05 indicated superiority in favor of treatment group with highest response; Odds Ratio (OR) = 1.51, 95% CI 2-sided [1.20 to 1.90]

29. Secondary Outcome: Percentage of Participants With Zero Incontinence Episodes Postbaseline
Description: Incontinence was defined as any involuntary leakage of urine.
Time Frame: Weeks 4, 8 and 12
Population: LOCF was used for EoT. The analysis population consisted of the FAS with data available at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Combination (Solifenacin + Mirabegron) | Solifenacin 5 mg | Solifenacin 10 mg
Number analyzed (Participants) | 707 | 705 | 698
percentage of participants
  Week 4: number analyzed (Participants) | 690 | 690 | 679
  Week 4 | 23.5 | 20.0 | 22.1
  Week 8: number analyzed (Participants) | 661 | 674 | 673
  Week 8 | 40.4 | 31.6 | 34.3
  Week 12: number analyzed (Participants) | 653 | 645 | 664
  Week 12 | 47.3 | 39.5 | 40.7
  EoT: number analyzed (Participants) | 706 | 704 | 697
  EoT | 46.0 | 37.9 | 40.2
Statistical Analysis 1: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 28, analysis 1]; Test type: Superiority; p = 0.119, Regression, Logistic — p<0.05 indicated superiority in favor of treatment group with highest response; Odds Ratio (OR) = 1.24, 95% CI 2-sided [0.95 to 1.63]
Statistical Analysis 2: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 28, analysis 2]; Test type: Superiority; p < 0.001, Regression, Logistic — p<0.05 indicated superiority in favor of treatment group with highest response; Odds Ratio (OR) = 1.56, 95% CI 2-sided [1.23 to 1.98]
Statistical Analysis 3: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 28, analysis 3]; Test type: Superiority; p = 0.002, Regression, Logistic — p<0.05 indicated superiority in favor of treatment group with highest response; Odds Ratio (OR) = 1.44, 95% CI 2-sided [1.14 to 1.82]
Statistical Analysis 4: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 28, analysis 4]; Test type: Superiority; p = 0.001, Regression, Logistic — p<0.05 indicated superiority in favor of treatment group with highest response; Odds Ratio (OR) = 1.47, 95% CI 2-sided [1.17 to 1.84]

30. Secondary Outcome: Percentage of Participants With a Mean of at Least 8 Micturitions Per 24 Hours at Baseline and Less Than 8 Micturitions Per 24 Hours Postbaseline
Description: Micturitions were defined as voluntary urinations (excluding incontinence only episodes).
Time Frame: Weeks 4, 8 and 12
Population: LOCF was used for EoT. The analysis population consisted of the FAS with data available at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Combination (Solifenacin + Mirabegron) | Solifenacin 5 mg | Solifenacin 10 mg
Number analyzed (Participants) | 707 | 705 | 698
percentage of participants
  Week 4: number analyzed (Participants) | 690 | 690 | 679
  Week 4 | 21.0 | 18.7 | 20.2
  Week 8: number analyzed (Participants) | 661 | 674 | 673
  Week 8 | 28.1 | 22.4 | 26.3
  Week 12: number analyzed (Participants) | 653 | 645 | 664
  Week 12 | 31.4 | 24.8 | 28.0
  EoT: number analyzed (Participants) | 706 | 704 | 697
  EoT | 30.2 | 25.0 | 27.7
Statistical Analysis 1: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 28, analysis 1]; Test type: Superiority; p = 0.305, Regression, Logistic — p<0.05 indicated superiority in favor of treatment group with highest response; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.88 to 1.50]
Statistical Analysis 2: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 28, analysis 2]; Test type: Superiority; p = 0.014, Regression, Logistic — p<0.05 indicated superiority in favor of treatment group with highest response; Odds Ratio (OR) = 1.37, 95% CI 2-sided [1.06 to 1.76]
Statistical Analysis 3: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 28, analysis 3]; Test type: Superiority; p = 0.012, Regression, Logistic — p<0.05 indicated superiority in favor of treatment group with highest response; Odds Ratio (OR) = 1.37, 95% CI 2-sided [1.07 to 1.76]
Statistical Analysis 4: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 28, analysis 4]; Test type: Superiority; p = 0.036, Regression, Logistic — p<0.05 indicated superiority in favor of treatment group with highest response; Odds Ratio (OR) = 1.29, 95% CI 2-sided [1.02 to 1.64]

31. Secondary Outcome: Percentage of Participants With at Least a 10-Point Improvement From Baseline in OAB-q Symptom Bother Score
Description: as for outcome 19
Time Frame: Weeks 4, 8 and 12
Population: LOCF was used for EoT. The analysis population consisted of the FAS with data available at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Combination (Solifenacin + Mirabegron) | Solifenacin 5 mg | Solifenacin 10 mg
Number analyzed (Participants) | 707 | 705 | 698
percentage of participants
  Week 4: number analyzed (Participants) | 682 | 677 | 669
  Week 4 | 67.9 | 58.2 | 61.9
  Week 8: number analyzed (Participants) | 670 | 660 | 658
  Week 8 | 77.2 | 66.4 | 69.1
  Week 12: number analyzed (Participants) | 644 | 641 | 647
  Week 12 | 83.5 | 72.1 | 75.4
  EoT: number analyzed (Participants) | 694 | 683 | 676
  EoT | 81.7 | 71.7 | 74.6
Statistical Analysis 1: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 28, analysis 1]; Test type: Superiority; p = 0.001, Regression, Logistic — p<0.05 indicated superiority in favor of treatment group with highest response; Odds Ratio (OR) = 1.49, 95% CI 2-sided [1.18 to 1.88]
Statistical Analysis 2: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 28, analysis 2]; Test type: Superiority; p < 0.001, Regression, Logistic — p<0.05 indicated superiority in favor of treatment group with highest response; Odds Ratio (OR) = 1.69, 95% CI 2-sided [1.31 to 2.18]
Statistical Analysis 3: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 28, analysis 3]; Test type: Superiority; p < 0.001, Regression, Logistic — p<0.05 indicated superiority in favor of treatment group with highest response; Odds Ratio (OR) = 1.96, 95% CI 2-sided [1.47 to 2.61]
Statistical Analysis 4: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 28, analysis 4]; Test type: Superiority; p < 0.001, Regression, Logistic — p<0.05 indicated superiority in favor of treatment group with highest response; Odds Ratio (OR) = 1.75, 95% CI 2-sided [1.34 to 2.30]

32. Secondary Outcome: Percentage of Participants With at Least a 10-Point Improvement From Baseline in HRQL Total Score
Description: HRQL subscales (coping, concern, sleep and social) and total score range from 0 (worst quality of life) to 100 (best quality of life).
Time Frame: Weeks 4, 8 and 12
Population: LOCF was used for EoT. The analysis population consisted of the FAS with data available at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Combination (Solifenacin + Mirabegron) | Solifenacin 5 mg | Solifenacin 10 mg
Number analyzed (Participants) | 707 | 705 | 698
percentage of participants
  Week 4: number analyzed (Participants) | 682 | 677 | 669
  Week 4 | 52.6 | 44.5 | 48.1
  Week 8: number analyzed (Participants) | 670 | 660 | 658
  Week 8 | 63.6 | 54.8 | 53.8
  Week 12: number analyzed (Participants) | 644 | 641 | 647
  Week 12 | 70.5 | 60.8 | 60.4
  EoT: number analyzed (Participants) | 694 | 683 | 676
  EoT | 68.6 | 60.6 | 60.1
Statistical Analysis 1: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 28, analysis 1]; Test type: Superiority; p = 0.003, Regression, Logistic — p<0.05 indicates superiority in favor of treatment group with highest response; Odds Ratio (OR) = 1.44, 95% CI 2-sided [1.14 to 1.82]
Statistical Analysis 2: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 28, analysis 2]; Test type: Superiority; p = 0.001, Regression, Logistic — p<0.05 indicates superiority in favor of treatment group with highest response; Odds Ratio (OR) = 1.51, 95% CI 2-sided [1.18 to 1.93]
Statistical Analysis 3: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 28, analysis 3]; Test type: Superiority; p < 0.001, Regression, Logistic — p<0.05 indicates superiority in favor of treatment group with highest response; Odds Ratio (OR) = 1.64, 95% CI 2-sided [1.27 to 2.13]
Statistical Analysis 4: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 28, analysis 4]; Test type: Superiority; p = 0.001, Regression, Logistic — p<0.05 indicates superiority in favor of treatment group with highest response; Odds Ratio (OR) = 1.50, 95% CI 2-sided [1.17 to 1.91]

33. Secondary Outcome: Percentage of Participants With at Least a 1-Point Improvement From Baseline in PPBC
Description: The PPBC was a validated, global assessment tool using a 6-point Likert scale on which participants rated their subjective impression of their current bladder condition.
Time Frame: Weeks 4, 8 and 12
Population: LOCF was used for EoT. The analysis population consisted of the FAS with data available at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Combination (Solifenacin + Mirabegron) | Solifenacin 5 mg | Solifenacin 10 mg
Number analyzed (Participants) | 707 | 705 | 698
percentage of participants
  Week 4: number analyzed (Participants) | 687 | 685 | 677
  Week 4 | 61.1 | 52.1 | 56.3
  Week 8: number analyzed (Participants) | 673 | 667 | 669
  Week 8 | 70.1 | 62.1 | 64.6
  Week 12: number analyzed (Participants) | 647 | 648 | 655
  Week 12 | 77.9 | 70.4 | 72.7
  EoT: number analyzed (Participants) | 697 | 688 | 683
  EoT | 76.5 | 69.5 | 71.9
Statistical Analysis 1: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 28, analysis 1]; Test type: Superiority; p = 0.003, Regression, Logistic — p<0.05 indicated superiority in favor of treatment group with highest response; Odds Ratio (OR) = 1.42, 95% CI 2-sided [1.13 to 1.79]
Statistical Analysis 2: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 28, analysis 2]; Test type: Superiority; p = 0.004, Regression, Logistic — p<0.05 indicated superiority in favor of treatment group with highest response; Odds Ratio (OR) = 1.44, 95% CI 2-sided [1.12 to 1.84]
Statistical Analysis 3: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 28, analysis 3]; Test type: Superiority; p = 0.003, Regression, Logistic — p<0.05 indicated superiority in favor of treatment group with highest response; Odds Ratio (OR) = 1.50, 95% CI 2-sided [1.15 to 1.96]
Statistical Analysis 4: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 28, analysis 4]; Test type: Superiority; p = 0.006, Regression, Logistic — p<0.05 indicated superiority in favor of treatment group with highest response; Odds Ratio (OR) = 1.43, 95% CI 2-sided [1.11 to 1.84]

34. Secondary Outcome: Percentage of Participants With Major (at Least 2-Point) Improvement From Baseline in PPBC
Description: as for outcome 33
Time Frame: Weeks 4, 8 and 12
Population: LOCF was used for EoT. The analysis population consisted of the FAS with data available at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Combination (Solifenacin + Mirabegron) | Solifenacin 5 mg | Solifenacin 10 mg
Number analyzed (Participants) | 707 | 705 | 698
percentage of participants
  Week 4: number analyzed (Participants) | 687 | 685 | 677
  Week 4 | 26.6 | 21.6 | 21.6
  Week 8: number analyzed (Participants) | 673 | 667 | 669
  Week 8 | 39.5 | 31.5 | 31.8
  Week 12: number analyzed (Participants) | 647 | 648 | 655
  Week 12 | 51.8 | 39.8 | 43.8
  EoT: number analyzed (Participants) | 697 | 688 | 683
  EoT | 49.8 | 39.1 | 43.2
Statistical Analysis 1: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 28, analysis 1]; Test type: Superiority; p = 0.065, Regression, Logistic; Odds Ratio (OR) = 1.28, 95% CI 2-sided [0.99 to 1.66]
Statistical Analysis 2: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 28, analysis 2]; Test type: Superiority; p = 0.004, Regression, Logistic; Odds Ratio (OR) = 1.41, 95% CI 2-sided [1.11 to 1.79]
Statistical Analysis 3: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 28, analysis 3]; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 1.64, 95% CI 2-sided [1.30 to 2.07]
Statistical Analysis 4: Comparison: Combination (Solifenacin + Mirabegron) vs Solifenacin 5 mg; [analysis description as in outcome 28, analysis 4]; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 1.55, 95% CI 2-sided [1.24 to 1.94]

35. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: AE was defined as any untoward medical occurrence in a participant administered a study drug or has undergone study procedures & which does not necessarily have a causal relationship with this treatment. Treatment-Emergent Adverse Event (TEAE) referred to an adverse event which started or worsened in the period from first double-blind medication intake until 30 days after the last double-blind medication intake.
Time Frame: From first dose of double blind treatment until 30 days after last dose (up to 16 weeks)
Population: The analysis population consisted of the Safety Analysis Set, the SAF comprised all randomized participants who received at least 1 dose of double-blind treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Combination (Solifenacin + Mirabegron) | Solifenacin 5 mg | Solifenacin 10 mg
Number analyzed (Participants) | 725 | 728 | 719
Participants
  AEs | 260 | 241 | 283
  Drug-related AEs | 141 | 125 | 161
  Serious Adverse Events (SAEs) | 13 | 10 | 15
  Drug-related SAEs | 1 | 0 | 3
  AEs Leading to Perm. Disc. of Study Drug | 11 | 11 | 11
  Drug-related AEs Leading to Perm. Disc. of Drug | 9 | 10 | 9
  Deaths | 0 | 0 | 0

36. Secondary Outcome: Change From Baseline in Post Void Residual (PVR) Volume
Description: PVR Volume was assessed by bladder scan.
Time Frame: Baseline and weeks 4, 8 & 12
Population: The analysis population consisted of the SAF with data available at each time point.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Combination (Solifenacin + Mirabegron) | Solifenacin 5 mg | Solifenacin 10 mg
Number analyzed (Participants) | 725 | 728 | 719
mL
  Week 4: number analyzed (Participants) | 705 | 712 | 704
  Week 4 | 1.545 (40.313) | 2.821 (38.588) | 7.308 (72.122)
  Week 8: number analyzed (Participants) | 683 | 694 | 690
  Week 8 | 2.245 (38.347) | 1.117 (36.470) | 7.232 (60.096)
  Week 12: number analyzed (Participants) | 669 | 680 | 681
  Week 12 | 6.356 (51.067) | 2.337 (42.147) | 6.552 (48.505)
  EoT: number analyzed (Participants) | 706 | 713 | 707
  EoT | 5.478 (51.595) | 3.046 (43.499) | 7.354 (54.121)

ADVERSE EVENTS:
Time Frame: From first dose of double blind treatment until 30 days after last dose (up to 16 weeks)
Description: Population consisted of the SAF. An AE was defined as any untoward medical occurrence in a participant administered a study drug or who had undergone study procedures and did not necessarily have a causal relationship with this treatment.
Arm/Group | Combination (Solifenacin + Mirabegron) | Solifenacin 5 mg | Solifenacin 10 mg
Serious Adverse Events (participants affected / at risk) | 13/725 | 10/728 | 15/719
Other Adverse Events (participants affected / at risk) | 43/725 | 41/728 | 68/719
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination (Solifenacin + Mirabegron) (N=725) | Solifenacin 5 mg (N=728) | Solifenacin 10 mg (N=719)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Adhesion (General disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Encephalitis herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Arteriogram coronary normal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Arthroscopy (Investigations) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Colonoscopy (Investigations) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cervix haemorrhage uterine (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Joint resurfacing surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Skin neoplasm excision (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination (Solifenacin + Mirabegron) (N=725) | Solifenacin 5 mg (N=728) | Solifenacin 10 mg (N=719)
Dry mouth (Gastrointestinal disorders) | 43 (44) | 41 (44) | 68 (70)

LIMITATIONS AND CAVEATS:
One participant was randomized to the Combination arm, but actually received Solifenacin 10 mg. In terms of actual treatment received, the participant was allocated to the solifenacin 10 mg arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI shall provide sponsor with a copy of proposed publication/presentation for review and comment at least 30 days prior to submission for publication/presentation. The sponsor can delay communications regarding trial results for an additional 90 days from the time submitted to the sponsor for review. The sponsor can require changes to the communication and can extend the delay.